CLINICAL TRIAL: NCT00256750
Title: Belatacept Evaluation of Nephroprotection and Efficacy as First-line Immunosuppression Trial (BENEFIT)
Brief Title: Belatacept Evaluation of Nephroprotection and Efficacy as First-line Immunosuppression (BENEFIT)
Acronym: BENEFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM103-008; NCT00432497 (obsolete NCT alias)
Record Dates: First submitted 2005-11-15; First posted 2005-11-22 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Transplantation; Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cyclosporine (CsA) (Active Comparator)
  Interventions: Drug: Cyclosporine (CsA)
- Belatacept LI (less intensive) (Experimental)
  Interventions: Drug: Belatacept LI (less intensive)
- Belatacept MI (more intensive) (Experimental)
  Interventions: Drug: Belatacept MI (more intensive)

INTERVENTIONS:
Drug: Cyclosporine (CsA) — tablet, oral, 1st month target: 150-300 ng/mL, after 1st month target: 100-250 ng/mL, daily, 36 months (ST), 100-250 ng/mL, daily, 24 months (LT)
  Arms: Cyclosporine (CsA)
Drug: Belatacept LI (less intensive) — solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 8 and 12, then 5 mg/kg every 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
  Arms: Belatacept LI (less intensive)
Drug: Belatacept MI (more intensive) — solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 6, 8, 10,12, 16, 20, and 24, then 5 mg/kg every 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
  Arms: Belatacept MI (more intensive)

SUMMARY:
The purpose of this study is to learn if Belatacept can provide protection from organ rejection following kidney transplantation while avoiding some of the toxic effects of standard immunosuppressive medications such as kidney damage. Effects on kidney function and patient survival as well as drug safety will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a recipient of a living donor or deceased donor kidney transplant.
* Male or Female, 18 or older

Exclusion Criteria:

* First time recipient, PRA >- 50% or for retransplantation PRA >- 30%.
* If retransplantation, previous graft loss cannot be due to acute rejection.
* Positive cross match.
* Subject receiving extended criteria donor (ECD) organ
* For Long-term extension study-Subjects who have completed three years of study treatment (through Week 156)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (102):
- United States (34):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center-Transplantation Institu, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Institute Of Renal Research, San Diego, California
  - University Of California San Francisco Medical Center, San Francisco, California
  - University Of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University School Of Medicine-Yale New Haven Hospital, New Haven, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Medical College Of Georgia, Augusta, Georgia
  - University Of Chicago Hospitals, Chicago, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Indiana
  - University Of Kentucky, Lexington, Kentucky
  - Maine Tranplant Program, Portland, Maine
  - Western New England Renal & Transplant Associates, Pc, Springfield, Massachusetts
  - Henry Ford Hospital, Transplant Institute, Detriot, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Recanati/Miller Transplantation Institute, New York, New York
  - Columbia University College Of Physicians & Surgeons, New York, New York
  - University Of Rochester Medical Center, Rochester, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Div Of Multi-Organ Trans, Hepato-Biliary-Pancreatic Surgery, Philadelphia, Pennsylvania
  - Musc, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Inova Transplant Center, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Sacred Heart Medical Ctr Providence Medical Research Ctr, Spokane, Washington
  - University Of Wisconsin, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (6):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Cordoba, Crd, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
- Australia (4):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Adelaide, South Australia
  - Local Institution, Parkville, Victoria
- Austria (2):
  - Local Institution, Innsbuck
  - Local Institution, Vienna
- Belgium (2):
  - Local Institution, Ghent
  - Local Institution, Leuven
- Brazil (6):
  - Local Institution, Rio de Janeiro / Rj, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre/rs, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Sao Paulo/sp, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Montreal, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Prague, Czechia
- France (7):
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Toulouse
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Hanover
- Local Institution, Szeged, Hungary
- India (9):
  - Local Institution, Gujarat, Ahmedabad
  - Local Institution, Chandigarh, Chandigarh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Nadiād, Gujarat
  - Local Institution, Kochi, Kerala
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Chennai
  - Local Institution, Lucknow
  - Local Institution, New Delhi
- Local Institution, Petah Tikva, Israel
- Italy (3):
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Roma
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
- Poland (2):
  - Local Institution, Poznan
  - Local Institution, Szczecin
- South Africa (3):
  - Local Institution, Observatory, Cape Town
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
- Local Institution, Gothenburg, Sweden
- Switzerland (2):
  - Local Institution, Bern
  - Local Institution, Zurich
- Local Institution, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Vincenti F, Rostaing L, Grinyo J, Rice K, Steinberg S, Gaite L, Moal MC, Mondragon-Ramirez GA, Kothari J, Polinsky MS, Meier-Kriesche HU, Munier S, Larsen CP. Belatacept and Long-Term Outcomes in Kidney Transplantation. N Engl J Med. 2016 Jan 28;374(4):333-43. doi: 10.1056/NEJMoa1506027. PMID 26816011
- [Derived] Dobbels F, Wong S, Min Y, Sam J, Kalsekar A. Beneficial effect of belatacept on health-related quality of life and perceived side effects: results from the BENEFIT and BENEFIT-EXT trials. Transplantation. 2014 Nov 15;98(9):960-8. doi: 10.1097/TP.0000000000000159. PMID 24831918
- [Derived] Vincenti F, Larsen CP, Alberu J, Bresnahan B, Garcia VD, Kothari J, Lang P, Urrea EM, Massari P, Mondragon-Ramirez G, Reyes-Acevedo R, Rice K, Rostaing L, Steinberg S, Xing J, Agarwal M, Harler MB, Charpentier B. Three-year outcomes from BENEFIT, a randomized, active-controlled, parallel-group study in adult kidney transplant recipients. Am J Transplant. 2012 Jan;12(1):210-7. doi: 10.1111/j.1600-6143.2011.03785.x. Epub 2011 Oct 12. PMID 21992533
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 738 participants enrolled, 686 randomized. Reasons for non-randomization include 5 participants withdrew consent, 1 lost to follow-up, 34 no longer met study criteria, and 12 for other non-listed reasons. 666 participants randomized, but not transplanted. 20 not transplanted; 10, 4, 6 in the CsA, Belatacept LI, Belatacept MI, respectively.
Groups:
- Cyclosporine: Cyclosporine (CsA): tablet, oral
  1st month target: 150-300 nanogram/meter (ng/m) After 1st month target: 100-250 nanogram/milliliter (ng/mL), daily, 36 months (short term = ST), 100-250 ng/mL, daily, 24 months (long term = LT)
- Belatacept LI: Belatacept LI (less intensive): solution, intravenous (IV), 10 milligrams/kilogram (mg/kg): Days 1 and 5, Weeks 2, 4, 8 and 12, then 5 mg/kg every (q) 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
- Belatacept MI: Belatacept MI (more intensive): solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 6, 8, 10,12, 16, 20, and 24, then 5 milligrams/kilogram (mg/kg) every 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
Period: Transplanted Pre-Treatment
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Started | 221 | 226 | 219
Completed | 215 | 226 | 219
Not Completed | 6 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Other | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: Post-Transplant Treated (12 Months)
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Started | 215 | 226 | 219
Completed | 174 | 183 | 173
Not Completed | 41 | 43 | 46
Not completed — Adverse Event | 20 | 12 | 8
Not completed — Death | 3 | 2 | 4
Not completed — Lack of Efficacy | 10 | 22 | 27
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 5 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 5
Not completed — Protocol Violation | 2 | 0 | 0
Period: Post-Transplant Treated (24 Months)
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Started | 174 | 183 | 173
Completed | 153 | 176 | 164
Not Completed | 21 | 7 | 9
Not completed — Adverse Event | 7 | 3 | 6
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Lack of Efficacy | 4 | 3 | 2
Not completed — Other | 2 | 0 | 1
Period: Post-Transplant Treated (36 Months)
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Started | 153 | 176 | 164
Completed | 143 | 170 | 158
Not Completed | 10 | 6 | 6
Not completed — Adverse Event | 5 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Death | 0 | 2 | 1
Not completed — Subject no longer meets study criteria | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Other | 0 | 1 | 1
Period: Long Term Extension (LTE; 84 Months)
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Started | 136 (Participants on drug through month 36 eligible to enroll in LTE; 2 ineligible, 5 withdrew or refused) | 166 (Participants on drug through month 36 were eligible to enroll in LTE; 4 withdrew or refused.) | 155 (Participants on drug through month 36 were eligible to enroll in LTE; 3 withdrew or refused.)
Completed | 89 | 136 | 127
Not Completed | 47 | 30 | 28
Not completed — Adverse Event | 13 | 11 | 14
Not completed — Withdrawal by Subject | 5 | 4 | 1
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Death | 9 | 4 | 4
Not completed — Lack of Efficacy | 6 | 3 | 0
Not completed — Poor/Non-compliance | 4 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 2
Not completed — Administrative Reason By Sponsor | 1 | 1 | 0
Not completed — Other | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of transplant recipients: All randomized and transplanted participants, intent to treat (ITT) population
Groups:
- Belatacept MI: Belatacept MI (more intensive): solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 6, 8, 10,12, 16, 20, and 24, then 5 mg/kg every 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI | Total
Number analyzed (Participants) | 221 | 226 | 219 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.3) | 42.6 (13.4) | 43.6 (14.6) | 43.2 (14.1)
Age, Customized [Number; unit: participants]
  Between 18 and 45 years: | 110 | 124 | 111 | 345
  Between 46 and 65 years: | 101 | 93 | 93 | 287
  > 65 years: | 10 | 9 | 15 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 80 | 68 | 204
  Male | 165 | 146 | 151 | 462
Previous Number of Transplant [Number; unit: participants]
  0 | 208 | 218 | 210 | 636
  1 | 9 | 5 | 5 | 19
  2 | 0 | 0 | 1 | 1
  Missing | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Surviving With a Functioning Graft by Month 12
Description: Graft loss was defined as either functional loss or physical loss (nephrectomy). Functional loss was defined as a sustained level of serum creatinine (SCr) ≥ 6.0 milligrams per deciliter (mg/dL) or 530 micromolar per liter (μmol/L) as determined by the central laboratory for ≥ 4 weeks or ≥ 56 consecutive days of dialysis or impairment of renal function to such a degree that the participant underwent retransplant.
Time Frame: Day 1 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 92.8 [89.3 to 96.2] | 96.5 [94.1 to 98.9] | 95.4 [92.7 to 98.2]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 10% for the co-primary endpoint of participant and graft survival was used. Determination of a margin for non-inferiority based on 'preservation of benefit' is not feasible, given the low rate of patient death and/or graft loss in the first year post-transplantation, and the absence of published, adequately sized, parallel-group trials with which to assess the effect of CsA on patient death and/or graft loss in the setting of MMF/steroids/basiliximab; Difference in Percent = 3.7, 97.3% CI 2-sided [-1.1 to 9.0]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Percent = 2.7, 97.3% CI 2-sided [-2.5 to 8.1] — If the lower bound of the CI (belatacept-CsA) was > -10%, then the corresponding belatacept regimen was considered non-inferior to CsA

2. Primary Outcome: Percent of Participants With a Composite of Measured Glomerular Filtration Rate (mGFR) Less Than 60 mL/Min/1.73 m^2 at Month 12 or With a Decrease in mGFR Greater Than or Equal to 10 mL/Min/1.73m^2 From Month 3 to Month 12
Description: Measured glomerular filtration rate (mGFR) is the direct measurement of renal function and was assessed by measurement of the clearance of a true glomerular filtration marker (non-radiolabeled iothalamate) using a validated procedure. A GFR of 60 mL/min/1.73 m^2 was used as the approximate equal of the threshold values of serum creatinine (SCr) of 1.5 mg/dL. A change in GFR of at least 10 mL/min/1.73 m^2 was used as the approximate change in SCr of at least 0.3 mg/dL. The change component of the composite renal endpoint was assessed from Month 3 to Month 12, since post-transplant renal function is largely stable by Month 3.
Time Frame: Month 12; Month 3 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 213 | 214 | 209
percentage of participants | 77.9 [72.4 to 83.5] | 54.2 [47.5 to 60.9] | 55.0 [48.3 to 61.8]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Superiority or Other; p < .0001, Chi-squared, Corrected; A continuity-corrected Chi-square test at significance level 0.027 was performed for the difference between the belatacept regimen and cyclosporine; Difference in Percent = -23.7, 97.3% CI 2-sided [-33.3 to -13.7]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; p < .0001, Chi-squared, Corrected; [statistical method as in outcome 2, analysis 1]; Difference in Percent = -22.9, 97.3% CI 2-sided [-32.6 to -12.9]

3. Primary Outcome: Percent of Participants Experiencing Acute Rejection (AR) Post-transplant by Month 12
Description: Acute rejection was defined as a clinico-pathological event requiring clinical evidence and biopsy confirmation. Clinical evidence was defined if either a or b was satisfied: a: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b: an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remains elevated within 14 days post-transplantation and clinical suspicion of acute rejection exists. Allograft biopsies were evaluated by a blinded central independent pathologist using Banff 97 working classification of kidney transplant pathology. Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. AR was defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Only the episode with the highest Banff grade for each participant was counted.
Time Frame: Day 1 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 7.2 [3.8 to 10.7] | 17.3 [12.3 to 22.2] | 21.9 [16.4 to 27.4]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Non-Inferiority or Equivalence — A 20% margin for non-inferiority was used and provides 99% power to ascertain that the upper bound of the 97.3% 2-sided confidence intervals for the absolute difference between each belatacept regimen and cyclosporine, assuming the true acute rejection rate by 12 months is 15% for all three regimens; Difference in Percent = 10.0, 97.3% CI 2-sided [3.3 to 17.1] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Non-Inferiority or Equivalence — A 20% margin for non-inferiority was used and provides 99% power to ascertain that the upper bound of the 97.3% 2-sided confidence intervals for the absolute difference between each belatacept regimen and cyclosporine, assuming the true acute rejection rate by 12 months is 15% for all three regimens. The 20% non-inferiority margin was not met in the belatacept MI group; Difference in Percent = 14.7, 97.3% CI 2-sided [7.5 to 22.2] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

4. Secondary Outcome: Mean Value of the Measured Glomerular Filtration Rate (mGFR)
Description: Measured glomerular filtration rate (mGFR) is the direct measurement of renal function and was assessed by measurement of the clearance of a true glomerular filtration marker (non-radiolabeled iothalamate) using a validated procedure. Missing mGRF assessments were imputed to assess renal function. The overall imputation strategy involved a primary imputation method (linear extrapolation and quartile method) followed by 2 secondary imputation methods (regression method and graded quartile method) to assess the robustness of conclusions obtained from the application of the primary imputation method. All imputation methods entailed replacing a missing value with a value drawn from a plausible distribution incorporating theoretical and observed aspects of the data. GFR was measured as mL/min/1.73 m^2.
Time Frame: Months 3, 12, 24
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 201 | 215 | 209
mL/min/1.73m^2
  Month 3 (n=201, 215, 209) | 51.9 (21.09) | 61.7 (25.43) | 59.9 (28.47)
  Month 12 (n=199, 206, 200) | 50.4 (18.71) | 63.4 (27.66) | 65.0 (30.02)
  Month 24 (n=185, 199, 192) | 50.5 (20.52) | 67.9 (29.90) | 65.0 (27.21)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Time Frame = Day 1 to Month 12; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis — To account for missing measured GFR due to graft loss or death, an ANOVA model on the ranks of measured GFR (with imputed missing values) at Months 12 with factor for randomization group was applied. Measured GFR missing were assigned the worst rank; Tests comparing a belatacept to CsA were based on the Kruskal-Wallis test (using a chi-square approximation of the distribution of the test statistic); Mean Difference (Final Values) = 13.0, 97.3% CI 2-sided [7.3 to 18.7] — Test were conducted at a level of 0.027 (2-sided)
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Time Frame = Day 1 to Month 12; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 14.6, 97.3% CI 2-sided [8.9 to 20.4] — Test were conducted at a level of 0.027 (2-sided)
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Time Frame = Day 1 to Month 24; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis — To account for missing measured GFR due to graft loss or death, an ANOVA model on the ranks of measured GFR (with imputed missing values) at Months 24 with factor for randomization group was applied. Measured GFR missing were assigned the worst rank; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 17.4, 97.3% CI 2-sided [11.5 to 23.4] — Test were conducted at a level of 0.027 (2-sided)
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Time Frame = Day 1 to Month 24; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis — [p-value comment as in outcome 4, analysis 3]; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = 14.5, 97.3% CI 2-sided [8.5 to 20.5] — Test were conducted at a level of 0.027 (2-sided)

5. Secondary Outcome: Percent of Participants With Prevalence of Chronic Allograft Nephropathy (CAN) at Month 12
Description: Prevalence of CAN = if participant met any of the following conditions: a: CAN observed in a biopsy either prior to 12 months (including baseline biopsy) or first post 12 months biopsy; b: participant had graft loss during the first year post transplant; c: no biopsy was available post 12 months and CAN not observed in biopsies prior to 12 months, but the measured GFR from Month 3 to Month 12 decreased at least 10 mL/min/1.73m^2; d: no biopsy available either prior to or post 12 months, and the measured GFR (incorporated missing data imputation) from Month 3 to Month 12 decreased at least 10 mL/min/1.73m^2. CAN = All allograft biopsies evaluated for presence and severity of CAN by a blinded central independent pathologist using Banff 97 working classification of kidney transplant pathology. Onset of CAN determined by the biopsy date when it was observed.
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component; Any participant not meeting CAN criteria and who has no biopsy either prior to or post 12 months and no GFR assessment (either measured or calculated) available were excluded from the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 219 | 226 | 219
percentage of participants | 32.4 [26.2 to 38.6] | 23.9 [18.3 to 29.5] | 18.3 [13.1 to 23.4]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Non-Inferiority or Equivalence — Test of superiority using DerSimonian-Laird statistic at 0.027 level of significance; p = 0.0581, Chi-squared, Corrected; A continuity corrected chi-square test at a significance level of 0.027 was performed; Difference in Percent = -8.5, 97.3% CI 2-sided [-17.9 to 0.9]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Non-Inferiority or Equivalence — Test of superiority using DerSimonian-Laird statistic at 0.027 level of significance; p = 0.0010, Chi-squared, Corrected; A continuity corrected chi-square test at a significance level of 0.027 was performed; Difference in Percent = -14.2, 97.3% CI 2-sided [-23.2 to -5.0]

6. Secondary Outcome: Number of Participants With Serious Adverse Events, Death, Discontinuation Due to Adverse Events by Month 84
Description: Adverse event (AE) defined: any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious adverse event (SAE) defined: a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Randomization to Month 84
Population: All randomized, transplanted, and treated participants from the original intent-to-treat (ITT) population who continued on assigned therapy into the long-term extension phase (ITT-LTE)
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 136 | 166 | 155
participants
  Deaths | 9 | 7 | 7
  SAEs | 107 | 113 | 117
  Discontinued due to SAEs | 5 | 8 | 6
  Discontinued due to AEs | 12 | 11 | 14

7. Secondary Outcome: Number of Participants With Adverse Events of Special Interest by Month 84
Description: Prospectively identified events of special interest which were a subset of all AEs, and were either SAEs or non-serious AEs, included the following categories: Serious Infections and Infestations, Thrombolic/embolic events, and Malignancy. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/ abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Time frame is from randomization to the event date, or to the last dose date+56, or to Month 84 (Day 2548), whichever is the earliest.
Time Frame: Randomization to Month 84
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 136 | 166 | 155
participants
  Malignancies | 22 | 16 | 20
  Cytomegalovirus (CMV) Infections | 19 | 24 | 20
  BK Polyoma Virus Infections | 6 | 10 | 15
  Herpes Virus Infections | 29 | 37 | 37
  Fungal Infections | 42 | 47 | 55
  Tuberculosis Infections | 2 | 1 | 5
  Central Nervous System (CNS) Infections | 0 | 0 | 1
  Pulmonary edema or Congestive Heart Failure | 12 | 4 | 5
  Auto-immune Events | 8 | 8 | 6

8. Secondary Outcome: Mean Blood Pressure at Month 84
Description: Blood pressure was measured in millimeters of mercury (mmHg). Blood pressure was measured soon after the participant arrived and sat quietly at rest for 10 minutes. 3 consecutive seated blood pressure readings were made at least 1 minute apart.
Time Frame: Month 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 136 | 166 | 155
mmHg
  Diastolic Blood Pressure (n=82, 125, 112) | 78.6 (11.03) | 75.8 (10.56) | 75.1 (10.15)
  Systolic Blood Pressure (n=82, 125, 112) | 129.0 (15.83) | 126.7 (18.17) | 126.0 (17.56)

9. Secondary Outcome: Number of Participants Meeting Marked Laboratory Abnormality Criteria Post-transplant by Month 36
Description: Upper limit of normal (ULN). Units per Liter (U/L). Cells per microliter (c/µL). Grams per deciliter (g/dL). Milligrams per deciliter (mg/dL).Cells per Liter (c/L). Milliequivalents/Liter (mEq/L).
  Hemoglobin (low): <8.0 g/dL; Platelet count: <50*10^9 c/L; Leukocytes: <2*10^3 c/µL; Alkaline phosphatase (ALP): >5.0*ULN U/L; Alanine aminotransferase (ALT): >5.0*ULN U/L; Asparate aminotransferase (AST): >5.0*ULN U/L; Bilirubin Total: >3.0*ULN mg/dL; Creatinine: >3.0*ULN mg/dL; Calcium Total: low if <7.0 mg/dL or high if >12.5 mg/dL; Bicarbonate: <11.0 mEq/L; Potassium serum: low if <3.0 mEq/L or high if >6.0 mEq/L; Magnesium serum: low is <0.8 mEq/L or high if >2.46 mEq/L; Sodium serum: low if <130.0 mEq/L or high if >155.0 mEq/L; Phosphorus inorganic: <2.0 mg/dL; Albumin: <2 g/dL; Uric acid: >10 mg/dL; Protein urine: >=3+
Time Frame: Baseline to Month 36
Population: All randomized, transplanted, and treated participants from the original intent-to-treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
participants
  Hemoglobin, low (n=213, 226, 219) | 26 | 25 | 27
  Platelet count, low (n=213, 226, 218) | 0 | 1 | 0
  Leukocytes, low (n=213, 226, 219) | 10 | 5 | 5
  Alkaline phosphatase, high (n=214, 226, 219) | 1 | 4 | 0
  Alanine aminotransferase, high (n=214, 226, 219) | 6 | 6 | 4
  Aspartate aminotransferase, high (n=214, 226, 219) | 2 | 3 | 3
  Bilirubin total, high (n=214, 226, 219) | 1 | 0 | 0
  Creatinine, high (n=213, 223, 219) | 48 | 50 | 52
  Calcium total, low (n=214, 226, 219) | 7 | 8 | 4
  Calcium total, high (n=214, 226, 219) | 0 | 1 | 0
  Bicarbonate, low (n=214, 226, 219) | 1 | 0 | 0
  Bicarbonate, high (n=214, 226, 219) | 0 | 0 | 0
  Potassium serum, low (n=213, 223, 219) | 4 | 13 | 12
  Potassium serum, high (n=213, 223, 219) | 13 | 9 | 4
  Magnessium serum, low (n=214, 225, 219) | 1 | 2 | 1
  Magnessium serum, high (n=214, 225, 219) | 9 | 12 | 14
  Sodium serum, low (n=214, 226, 219) | 21 | 8 | 9
  Sodium serum, high (n=214, 226, 219) | 0 | 1 | 0
  Phosphorus inorganic, low (n=213, 224, 219) | 75 | 100 | 112
  Albumin, low (n=214, 226, 219) | 0 | 0 | 0
  Uric acid, high (n=214, 226, 219) | 42 | 7 | 11
  Protein in urine, high (n=213, 224, 217) | 33 | 30 | 36

10. Secondary Outcome: Percent of Participants With Development of Anti-Donor HLA Positive Antibodies by Month 84
Description: Only participants who had non-missing test result for Class I or Class II anti-donor HLA antibodies were included in analysis and only participants who had at least one non-NA test result or finding were counted. This was a cumulative summary (excluding baseline) and once a participant was positive, that participant remained positive for the later time point. Acute rejection (AR) defined: a clinico-pathological event requiring clinical evidence and biopsy confirmation. Clinical evidence defined: if either a or b was satisfied: a: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b: an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remains elevated within 14 days post-transplantation and clinical suspicion of acute rejection exists. AR defined as allograft biopsies of Banff 97 classification Grade IA or greater (higher scores indicate more severe rejection). Evaluated by blinded central independent pathologist.
Time Frame: Randomization to Month 84
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 215 | 226 | 219
percentage of participants | 11.6 [7.34 to 15.91] | 3.1 [0.84 to 5.36] | 1.4 [0.28 to 3.95]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Percent treatment difference measured as Belatacept - LI minus Cyclosporine; Test type: Superiority or Other; Difference in Percent = -8.5, 97.3% CI 2-sided [-14.6 to -3.3] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Percent treatment difference measured as Belatacept - LI minus Cyclosporine; Test type: Superiority or Other; Difference in Percent = -10.3, 97.3% CI 2-sided [-16.1 to -5.1] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

11. Secondary Outcome: Mean Change of the Measured Glomerular Filtration Rate (mGFR) From Month 3 to Month 12 and From Month 3 to Month 24
Description: as for outcome 4
Time Frame: Month 3 to Month 12; Month 3 to Month 24
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 195 | 206 | 200
mL/min/1.73m^2
  Baseline (Month 3) to Month 12 (n=195, 206, 200) | -1.7 (21.58) | 1.2 (30.43) | 4.4 (31.10)
  Baseline (Month 3) to Month 24 (n=184, 199, 192) | -2.0 (25.23) | 5.3 (33.03) | 4.2 (30.96)

12. Secondary Outcome: Percent of Participants With a Decrease in Measured Glomerular Filtration Rate (mGFR) Greater Than or Equal to 10mL/Min/1.73m^2 From Month 3 to Month 12
Description: Measured glomerular filtration rate (mGFR) is the direct measurement of renal function and was assessed by measurement of the clearance of a true glomerular filtration marker (non-radiolabeled iothalamate) using a validated procedure. A change in GFR of at least 10 mL/min/1.73 m^2 was used as the approximate change in serum creatinine (SCr) of at least 0.3 mg/dL. The change component of the composite renal endpoint was assessed from Month 3 to Month 12, since post-transplant renal function is largely stable by Month 3. Month 3 = baseline
Time Frame: Month 3 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 213 | 214 | 209
percentage of participants | 28.2 [22.1 to 34.2] | 23.4 [17.7 to 29.0] | 23.0 [17.3 to 28.7]

13. Secondary Outcome: Percent of Participants With a Measured Glomerular Filtration Rate (mGFR) Less Than 60 mL/Min/1.73 m^2 at Month 12
Description: Measured glomerular filtration rate (mGFR) is the direct measurement of renal function and was assessed by measurement of the clearance of a true glomerular filtration marker (non-radiolabeled iothalamate) using a validated procedure. A GFR of 60 mL/min/1.73 m^2 was used as the approximate equal of the threshold values of serum creatinine (SCr) of 1.5 milligrams per deciliter (mg/dL).
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 213 | 214 | 209
percentage of participants | 67.6 [61.3 to 73.9] | 43 [36.4 to 49.6] | 43.5 [36.8 to 50.3]

14. Secondary Outcome: Mean Value of the Calculated Glomerular Filtration Rate (cGFR) With Imputation
Description: Calculated glomerular filtration rate (cGFR) was used to assess renal function (as measured by the estimated creatinine clearance) using the following modification of diet in renal disease (MDRD) formula: MDRD: GFR = 170 x [SCr/0.95]^(-0.999) x [Age]^(-0.176) x [0.762 if participant is female] x [1.180 if participant is black] x [BUN]^(-0.170) x [Alb]^(+0.318); Age in years; Alb = Albumin in g/dL; SCr = Serum creatinine in mg/dL; BUN = Blood urea nitrogen in mg/dL; cGFR = mL/min/1.73m2
Time Frame: Months 6, 12, 24, 36
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 199 | 201 | 201
mL/min/1.73 m^2
  Month 6 (n=189, 185, 170) | 48.8 (19.22) | 62.6 (20.41) | 62.4 (20.94)
  Month 12 (n=199, 200, 201) | 50.1 (21.06) | 65.4 (22.94) | 65.2 (23.51)
  Month 24 (n=182, 201, 191) | 47.9 (23.00) | 65.4 (25.22) | 65.5 (24.87)
  Month 36 (n=171, 190, 186) | 44.4 (23.58) | 65.8 (27.00) | 65.2 (26.31)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = 15.3, 97.3% CI 2-sided [10.3 to 20.3] — ANOVA model: GFR = treatment
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = 15.1, 97.3% CI 2-sided [10.1 to 20.1] — ANOVA model: GFR = treatment
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = 17.5, 97.3% CI 2-sided [12.0 to 23.1] — ANOVA model: GFR = treatment
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = 17.6, 97.3% CI 2-sided [12.0 to 23.3] — ANOVA model: GFR = treatment
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = 21.4, 97.3% CI 2-sided [15.4 to 27.4] — ANOVA model: GFR = treatment
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = 20.8, 97.3% CI 2-sided [14.8 to 26.9] — ANOVA model: GFR = treatment

15. Secondary Outcome: Mean Change in Calculated Glomerular Filtration Rate (cGFR) From Month 6 to Month 12
Description: Calculated glomerular filtration rate (cGFR) was used to assess renal function (as measured by the estimated creatinine clearance) using the following modification of diet in renal disease (MDRD) formula: MDRD: GFR = 170 x [SCr/0.95]^(-0.999) x [Age]^(-0.176) x [0.762 if participant is female] x [1.180 if participant is black] x [BUN]^(-0.170) x [Alb]^(+0.318); Age in years; Alb = Albumin in g/dL; SCr = Serum creatinine in mg/dL; BUN = Blood urea nitrogen in mg/dL; cGFR = mL/min/1.73m^2
Time Frame: Month 6 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Mean (Standard Deviation); unit: mL/Min/1.73 m^2
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 166 | 169 | 160
mL/Min/1.73 m^2 | 2.3 (10.09) | 4.7 (11.52) | 5.1 (11.37)

16. Secondary Outcome: Percent of Participants With Incidence of New Onset Diabetes Mellitus by Month 36
Description: The incidence of new onset diabetes mellitus defined as participants who developed diabetes mellitus after randomization and transplantation. Participants that did not have diabetes prior to randomization were determined to have new onset diabetes mellitus if (i) the participant received an anti-diabetic medication for a duration of at least 30 days or (ii) at least two fasting plasma glucose (FPG) tests indicate that FPG is >=126 mg/dL (7.0 mmol/L). New onset diabetes mellitus (NODM) = post-transplant diabetes mellitus (PTDM)
Time Frame: Week 4 post-transplantation to Month 36
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 162 | 168 | 156
percentage of participants
  Month 12 | 9.9 [5.3 to 14.5] | 4.2 [1.1 to 7.2] | 7.1 [3.0 to 11.1]
  Month 24 | 10.5 [5.8 to 15.2] | 5.4 [2.0 to 8.8] | 8.3 [4.0 to 12.7]
  Month 36 | 11.1 [6.3 to 16.0] | 6.5 [2.8 to 10.3] | 10.3 [5.5 to 15.0]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; p = 0.0687, Chi-squared — Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -5.7, 97.3% CI 2-sided [-12.6 to 0.5]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 12; Test type: Superiority or Other; p = 0.4825, Chi-squared — Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -2.8, 97.3% CI 2-sided [-10.2 to 4.4]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Month 24; Test type: Superiority or Other; p = 0.1267, Chi-squared — Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -5.1, 97.3% CI 2-sided [-12.3 to 1.5]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Month 24; Test type: Superiority or Other; p = 0.6405, Chi-squared — Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -2.2, 97.3% CI 2-sided [-9.8 to 5.4]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Month 36; Test type: Superiority or Other; p = 0.2043, Chi-squared; Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -4.6, 97.3% CI 2-sided [-12.0 to 2.5]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Month 36; Test type: Superiority or Other; p = 0.9481, Chi-squared — Normal approximation is used if N>=5 in both arms. Otherwise, exact method is used; Difference in Percent = -0.9, 97.3% CI 2-sided [-8.8 to 7.1]

17. Secondary Outcome: Percent of Participants Using At Least One Anti-Hypertensive Medication to Control Hypertension at Month 36
Description: This analysis was based on all participants who had been followed up at least 1092 days after transplantation. Hypertension was defined in according to the Seventh Report of the Joint National Committee on the Prevention, Detection, Evaluation, and Treatment of High Blood Pressure for participants with chronic kidney disease. This definition was based upon SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg. In addition, all participants who had a SBP < 130 mm Hg and a DBP < 80 mm Hg who received an antihypertensive medication(s) for the indication of hypertension or with a medical history of hypertension were included in this definition. Systolic blood pressure = SBP; Diastolic blood pressure = DBP
Time Frame: Month 36
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 182 | 199 | 192
percentage of participants | 92.9 [89.12 to 96.60] | 81.9 [76.56 to 87.36] | 83.9 [78.65 to 89.06]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Superiority or Other; p = 0.0002, Chi-squared; Odds Ratio (OR) = 0.5, 97.3% CI 2-sided [0.31 to 0.74] — Odds ratio is estimated by a cumulative logit model
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; p = 0.0092, Chi-squared; Odds Ratio, log = 0.6, 97.3% CI 2-sided [0.38 to 0.92] — Odds ratio is estimated by a cumulative logit model

18. Secondary Outcome: Percent of Participants With Incidence of Hypertension Post-Transplantation at Month 12
Description: The incidence of hypertension was defined as the proportion of participants who developed hypertension after randomization and transplantation. Specifically, the incidence of hypertension was assessed only after the Week 4 visit. This period allowed for adequate stabilization and resolution of transient changes. If participants received antihypertensive medication for the indication of hypertension at this (or later) time point, they were considered to have developed hypertension. Hypertension was defined according to the Seventh Report of the Joint National Committee on the Prevention, Detection, Evaluation, and Treatment of High Blood Pressure for subjects with chronic kidney disease. This definition was based upon SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg. Systolic blood pressure = SBP; Diastolic blood pressure = DBP
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 4 | 13 | 7
percentage of participants | 75.0 [19.4 to 99.4] | 53.8 [26.7 to 80.9] | 57.1 [18.4 to 90.1]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; Difference in Percent = -21.2, 97.3% CI 2-sided [-67.6 to 43.2] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 12; Test type: Superiority or Other; Difference in Percent = -17.9, 97.3% CI 2-sided [-72.3 to 52.2] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

19. Secondary Outcome: Percent of Participants With Prevalence of Hypertension Post-Transplantation at Month 12
Description: The prevalence of hypertension was defined as the proportion of participants at any given time who meet the definition of hypertension. Hypertension defined according to the Seventh Report of the Joint National Committee on the Prevention, Detection, Evaluation, and Treatment of High Blood Pressure for participants with chronic kidney disease. This definition is based upon SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg. Systolic blood pressure = SBP; Diastolic blood pressure = DBP
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 91.0 [87.17 to 94.73] | 89.8 [85.88 to 93.76] | 88.6 [84.37 to 92.80]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; Difference in Percent = -1.13, 97.3% CI 2-sided [-7.51 to 5.23] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 12; Test type: Superiority or Other; Difference in Percent = -2.37, 97.3% CI 2-sided [-9.01 to 4.15] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

20. Secondary Outcome: Mean Systolic Blood Pressure and Diastolic Blood Pressure
Description: as for outcome 8
Time Frame: Months 12, 24, 36
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 188 | 193 | 191
mmHg
  Systolic; Month 12 (n=188, 193, 191) | 138.7 (19.98) | 131.4 (16.54) | 132.7 (16.21)
  Diastolic; Month 12 (n=188, 193, 191) | 81.9 (11.10) | 78.7 (10.91) | 79.3 (11.54)
  Systolic; Month 24 (n=160, 185, 174) | 135.4 (19.71) | 130.5 (17.35) | 129.8 (16.84)
  Diastolic; Month 24 (n=160, 185, 174) | 80.3 (10.20) | 78.3 (10.51) | 77.8 (10.31)
  Systolic; Month 36 (n=145, 180, 166) | 133.5 (17.93) | 127.7 (16.48) | 126.0 (16.14)
  Diastolic; Month 36 (n=145, 180, 166) | 79.5 (9.16) | 76.6 (9.75) | 76.1 (11.20)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Systolic, Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = -7.3, 97.3% CI 2-sided [-11.4 to -3.3]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Systolic, Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = -6.0, 97.3% CI 2-sided [-10.1 to -2.0]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Diastolic, Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = -3.2, 97.3% CI 2-sided [-5.8 to -0.7]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Diastolic, Month 12; Test type: Superiority or Other; Mean Difference (Final Value) = -2.6, 97.3% CI 2-sided [-5.1 to 0.0]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Systolic, Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = -4.9, 97.3% CI 2-sided [-9.2 to -0.6]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Systolic, Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = -5.5, 97.3% CI 2-sided [-9.9 to -1.1]
Statistical Analysis 7: Comparison: Cyclosporine vs Belatacept LI; Diastolic, Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = -1.9, 97.3% CI 2-sided [-4.4 to 0.5]
Statistical Analysis 8: Comparison: Cyclosporine vs Belatacept MI; Diastolic, Month 24; Test type: Superiority or Other; Mean Difference (Final Value) = -2.4, 97.3% CI 2-sided [-5.0 to 0.1]
Statistical Analysis 9: Comparison: Cyclosporine vs Belatacept LI; Systolic, Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = -5.8, 97.3% CI 2-sided [-10.0 to -1.6]
Statistical Analysis 10: Comparison: Cyclosporine vs Belatacept MI; Systolic, Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = -7.5, 97.3% CI 2-sided [-11.7 to -3.3]
Statistical Analysis 11: Comparison: Cyclosporine vs Belatacept LI; Diastolic, Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = -2.9, 97.3% CI 2-sided [-5.4 to -0.4]
Statistical Analysis 12: Comparison: Cyclosporine vs Belatacept MI; Diastolic, Month 36; Test type: Superiority or Other; Mean Difference (Final Value) = -3.4, 97.3% CI 2-sided [-6.0 to -0.9]

21. Secondary Outcome: Percent of Participants at Baseline With Controlled Hypertension Post Transplantation by Month 12
Description: Controlled hypertension was defined as a SBP < 130 mm Hg and a DBP < 80 mm Hg while receiving an antihypertensive medication for the indication of hypertension or receiving an antihypertensive medication for another indication with a medical history of hypertension. Participants with a SBP < 130 mm Hg and a DBP < 80 mm Hg who were prescribed an antihypertensive medication(s) for an indication(s) other than hypertension (eg, beta blockers for migraine prophylaxis) with no medical history of hypertension were not considered to have either hypertension or controlled hypertension. Systolic blood pressure = SBP; Diastolic blood pressure = DBP
Time Frame: Day 1 to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with baseline hypertension
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 182 | 182 | 183
percentage of participants | 21.4 [15.5 to 27.4] | 28.6 [22.0 to 35.1] | 24.6 [18.4 to 30.8]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; At Month 12; Test type: Superiority or Other; Difference in Percent = 7.1, 97.3% CI 2-sided [-2.9 to 17.1] — A continuity-corrected Chi-square test at significance level 0.027 was performed for the difference between the belatacept regimen and cyclosporine
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; At Month 12; Test type: Superiority or Other; Difference in Percent = 3.2, 97.3% CI 2-sided [-6.6 to 12.9] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Percent of Participants With Prevalence of Controlled Hypertension at Month 12
Description: The prevalence of controlled hypertension was defined as the proportion of participants at any given time who met the definition of controlled hypertension. Controlled hypertension was defined as a SBP < 130 mm Hg and a DBP < 80 mm Hg while receiving an antihypertensive medication for the indication of hypertension or receiving an antihypertensive medication for another indication with a medical history of hypertension. Participants with a SBP < 130 mm Hg and a DBP < 80 mm Hg who were prescribed an antihypertensive medication(s) for an indication(s) other than hypertension (eg, beta blockers for migraine prophylaxis) with no medical history of hypertension were not considered to have either hypertension or controlled hypertension. Systolic blood pressure = SBP; Diastolic blood pressure = DBP
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 186 | 193 | 190
percentage of participants | 21.0 [15.12 to 26.82] | 28.0 [21.65 to 34.31] | 24.7 [18.60 to 30.87]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Superiority or Other; Difference in Percent = 7.01, 97.3% CI 2-sided [-2.79 to 16.71] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; Difference in Percent = 3.77, 97.3% CI 2-sided [-5.86 to 13.35] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: Percent of Non-dyslipidemic Participants With Incidence of Dyslipidemia Post-Transplantation by Month 12
Description: Incidence of dyslipidemia was defined as the proportion of participants who developed dyslipidemia after randomization and transplantation. Dyslipidemia was defined in accordance with recent guidelines from the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF-K/DOQI). Dyslipidemia = hypertriglyceridemia (TGs >= 500 milligrams/deciliter (mg/dL) [5.65 mmol/L]), hypercholesterolemia (LDL >= 100 mg/dL [2.59 mmol/L]), or elevated non-HDL (non-HDL >= 130 mg/dL [3.36 mmol/L]) in the presence of high TGs (TGs >= 200 mg/dL [2.26 mmol/L]). The TG = triglyceride; LDL = low density lipoprotein; HDL = high density lipoprotein; millimole/Liter (mmol/L). For 95% CI within each group, normal approximation is used if N >=5. Otherwise exact method is used.
Time Frame: Randomization to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 75 | 94 | 79
percentage of participants | 80.0 [70.9 to 89.1] | 63.8 [54.1 to 73.5] | 70.9 [60.9 to 80.9]

24. Secondary Outcome: Percent of Participants With Prevalence of Dyslipidemia at Month 12
Description: The prevalence of dyslipidemia was defined as the proportion of participants at any given time who met the definition of dyslipidemia. Dyslipidemia defined in accordance with recent guidelines from the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF-K/DOQI). Dyslipidemia defined as hypertriglyceridemia (TGs >= 500 milligrams/deciliter (mg/dL) [5.65 mmol/L]), hypercholesterolemia (LDL >= 100 mg/dL [2.59 mmol/L]), or elevated non-HDL (non-HDL >= 130 mg/dL [3.36 mmol/L]) in the presence of high TGs (TGs >= 200 mg/dL [2.26 mmol/L]). TG = triglyceride; LDL = low density lipoprotein; HDL = high density lipoprotein; millimole/Liter (mmol/L). For 95% CI within each group, normal approximation is used if N >=5. Otherwise exact method is used.
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 52.9 [46.4 to 59.5] | 44.7 [38.2 to 51.2] | 46.1 [39.5 to 52.7]

25. Secondary Outcome: Percent of Participants With Controlled Dyslipidemia at Month 12
Description: Prevalence of controlled dyslipidemia = the proportion of participants at any given time who met the stated definition of dyslipidemia. Dyslipidemia defined in accordance with recent guidelines from the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF-K/DOQI). Dyslipidemia defined as hypertriglyceridemia (TGs >= 500 milligrams/deciliter (mg/dL) [5.65 mmol/L]), hypercholesterolemia (LDL >= 100 mg/dL [2.59 mmol/L]), or elevated non-HDL (non-HDL >= 130 mg/dL [3.36 mmol/L]) in the presence of high TGs (TGs >= 200 mg/dL [2.26 mmol/L]). Controlled dyslipidemia defined as participants who received successful pharmacologic treatment for 1 of the above stated dyslipidemias, and their lipid values fell below the thresholds described. TG = triglyceride; LDL = low density lipoprotein; HDL = high density lipoprotein; millimole/Liter (mmol/L). For 95% CI within each group, normal approximation is used if N >=5. Otherwise exact method is used.
Time Frame: Month 12
Population: All randomized and transplanted participants, intent-to-treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 18.1 [13.0 to 23.2] | 15.5 [10.8 to 20.2] | 15.5 [10.7 to 20.3]

26. Secondary Outcome: Number of Participants With Antihyperlipidemic Medication by Intensity Level
Description: An intensity level was associated with the dose level of the statin based anti-hyperlipidemic agent. Any other agent (i.e., non-statin therapy) used as an antihyperlipidemic were considered Level I treatment intensity. Multiple daily dose levels during a period were averaged to compute the daily dose during that period. Level I = 20 mg fluvastatin (flu), 10 mg lovastatin (lova), 10 mg pravastatin (prav), 5-10 mg simvastatin (sim); Level II = 10 mg atorvastatin (atorv), 40 mg flu, 20 mg lova, 20 mg prav, 5 mg rosuvastatin (rosu), 20 mg sim, 10/10 vytorin; Level III = 20 mg atorv, 80 mg flu, 40 mg lova, 40 mg prav, 10 mg rosu, 40 mg sim, 10/20 vytorin; Level IV = 40 mg atorv, 80 mg lova, 80 mg prav, 20 mg rosu, 80 mg sim, 10/40 vytorin; Level V = 80 mg atorv, 40 mg rosu, 10/80 vytorin. Concomitant use of a statin and an agent of another class elevated the intensity level of the statin therapy by 1 level; therefore, an intensity level of greater than V was possible.
Time Frame: Month 36
Population: All randomized and transplanted participants that received at least one hyperlipidemic medication; Completer analysis is based on all participants who have been followed up at least 1092 days after transplantation.
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 103 | 92 | 92
participants
  Intensity Level I | 17 | 15 | 17
  Intensity Level II | 46 | 27 | 39
  Intensity Level III | 27 | 32 | 23
  Intensity Level IV | 8 | 16 | 9
  Intensity Level V | 4 | 1 | 4
  Intensity Level VI | 1 | 1 | 0

27. Secondary Outcome: Percent of Participants Using At Least One Anti-Hyperlipidemic Medication
Description: This analysis is based on all participants who were followed up at least 1092 days after transplantation.
Time Frame: Month 36
Population: All randomized and transplanted participants, intent-to-treat (ITT) population; Completer analysis is based on all participants who have been followed up at least 1092 days after transplantation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 182 | 199 | 192
percentage of participants | 56.6 [49.4 to 63.8] | 46.2 [39.3 to 53.2] | 47.9 [40.9 to 55.0]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Superiority or Other; Difference in Percent = -10.4, 97.3% CI 2-sided [-21.4 to 1.0]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; Difference in Percent = -8.7, 97.3% CI 2-sided [-19.9 to 2.7]

28. Secondary Outcome: Mean Value of Lipid Parameters
Description: Lipid parameters included total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, non-HDL cholesterol, and triglycerides (TGs).
Time Frame: Months 12, 24, 36
Population: All randomized and transplanted participants, intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 189 | 195 | 192
mg/dL
  non-HDL Cholesterol; Month 12 (n=189, 195, 192) | 144.1 (47.31) | 131.5 (38.18) | 131.7 (36.76)
  Total Cholesterol; Month 12 (n=189, 195, 192) | 191.5 (49.29) | 182.4 (39.78) | 181.3 (39.92)
  HDL Cholesterol; Month 12 (n=189, 195, 192) | 47.4 (13.33) | 50.8 (15.98) | 49.7 (15.69)
  LDL Cholesterol; Month 12 (n=187, 186, 183) | 107.3 (39.60) | 102.1 (33.40) | 100.8 (29.48)
  Triglyceride; Month 12 (n=187, 186, 183) | 184.6 (106.42) | 149.4 (87.25) | 155.0 (85.08)
  non-HDL Cholesterol; Month 24 (n=166, 190, 181) | 145.1 (39.52) | 126.7 (38.48) | 127.0 (36.76)
  Total Cholesterol; Month 24 (n=166, 190, 181) | 193.5 (40.23) | 175.3 (42.38) | 175.4 (40.03)
  HDL ; Month 24 (n=166, 190, 181) | 48.4 (13.74) | 48.6 (15.28) | 48.5 (14.92)
  LDL Cholesterol; Month 24 (n=164, 186, 168) | 109.1 (35.92) | 98.6 (33.71) | 96.5 (30.52)
  Triglyceride; Month 24 (n=164, 186, 168) | 179.5 (97.51) | 143.4 (88.97) | 151.2 (95.88)
  non-HDL Cholesterol; Month 36 (n=154, 184, 176) | 142.2 (43.19) | 122.4 (40.12) | 122.1 (38.78)
  Total Cholesterol; Month 36 (n=154, 184, 176) | 190.7 (45.28) | 171.3 (45.78) | 170.7 (43.26)
  HDL Cholesterol; Month 36 (n=154, 184, 176) | 48.5 (14.27) | 48.9 (15.37) | 48.6 (16.86)
  LDL Cholesterol; Month 36 (n=142, 170, 161) | 107.6 (37.66) | 96.7 (36.53) | 92.5 (33.78)
  Triglyceride; Month 36 (n=142, 170, 161) | 179.1 (97.07) | 132.7 (68.69) | 144.0 (81.48)

29. Secondary Outcome: Percent of Participants With Prevalence of Acute Rejection (AR) by Month 36
Description: Prevalence of AR = participants with the stated definition of AR at any given time. AR defined as a clinico-pathological event requiring clinical evidence and renal biopsy confirmation demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Only the episode with the highest Banff grade for each participant was counted. Clinical evidence = if either a or b was satisfied: a: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b: an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remains elevated within 14 days post-transplantation and clinical suspicion of acute rejection exists. Allograft biopsies were evaluated by a blinded central independent pathologist using Banff 97 working classification of kidney transplant pathology. Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants
  Month 6 (n=221, 226, 219) | 5.4 [2.4 to 8.4] | 16.8 [11.9 to 21.7] | 21.9 [16.4 to 27.4]
  Month 24 (n=221, 226, 219) | 9.0 [5.3 to 12.8] | 17.3 [12.3 to 22.2] | 24.2 [18.5 to 29.9]
  Month 36 (n=221, 226, 219) | 9.5 [5.6 to 13.4] | 17.3 [12.3 to 22.2] | 24.2 [18.5 to 29.9]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 11.4, 97.3% CI 2-sided [5.0 to 18.2] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 16.5, 97.3% CI 2-sided [9.6 to 23.8] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Month 24; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 8.2, 97.3% CI 2-sided [1.2 to 15.4] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Month 24; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 15.2, 97.3% CI 2-sided [7.5 to 23.0] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Month 36; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 7.8, 97.3% CI 2-sided [0.6 to 15.0] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Month 36; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in Percent = 14.7, 97.3% CI 2-sided [7.0 to 22.6] — For 97.3% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

30. Secondary Outcome: Number of Participants With Acute Rejection (AR) Post-transplant in Terms of Severity Using Banff Grades by Month 36
Description: Acute rejection was defined as a clinico-pathological event requiring clinical evidence and renal biopsy confirmation demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Clinical evidence defined: if either a or b was satisfied: a) an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b) an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remains elevated within 14 days post-transplantation and clinical suspicion of acute rejection exists. Allograft biopsies were evaluated by a blinded central independent pathologist using Banff 97 working classification of kidney transplant pathology. Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Only the episode with the highest Banff grade for each participant was counted.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
participants
  Mild Acute (IA); Month 6 | 1 | 4 | 7
  Mild Acute (IB); Month 6 | 5 | 9 | 3
  Moderate Acute (IIA); Month 6 | 5 | 14 | 16
  Moderate Acute (IIB); Month 6 | 1 | 10 | 20
  Severe Acute (III); Month 6 | 0 | 1 | 2
  Mild Acute (IA); Month 12 | 3 | 4 | 7
  Mild Acute (IB); Month 12 | 5 | 8 | 3
  Moderate Acute (IIA); Month 12 | 6 | 16 | 17
  Moderate Acute (IIB); Month 12 | 2 | 10 | 20
  Severe Acute (III); Month 12 | 0 | 1 | 2
  Mild Acute (IA); Month 24 | 4 | 4 | 7
  Mild Acute (IB); Month 24 | 7 | 8 | 3
  Moderate Acute (IIA); Month 24 | 6 | 16 | 18
  Moderate Acute (IIB); Month 24 | 3 | 10 | 22
  Severe Acute (III); Month 24 | 0 | 1 | 3
  Mild Acute (IA); Month 36 | 5 | 4 | 7
  Mild Acute (IB); Month 36 | 7 | 8 | 3
  Moderate Acute (IIA); Month 36 | 6 | 16 | 18
  Moderate Acute (IIB); Month 36 | 3 | 10 | 22
  Severe Acute (III); Month 36 | 0 | 1 | 3

31. Secondary Outcome: Percent of Participants Using Polyclonal Antilymphocyte Preparations for Impaired Renal Function and Anticipated Delayed Graft Function by Month 12
Description: A participant was considered to have delayed graft function (DGF), if treated with dialysis within the first week (Day 1 - 8) after transplantation. The use of polyclonal antilymphocyte preparations (LDT) was permitted only for participants randomized to cyclosporine (CsA) who experienced impaired renal allograft function and anticipated DGF following transplantation and were not permitted in belatacept-treated participants, except for the treatment of acute rejection. Participants treated with LDT began CsA at the discretion of the investigator by Day 7. LDT could also have been used in participants who met >= 1 of the following criteria, observed in the presence of a transplant artery and vein and no evidence of hydronephrosis by sonogram: Urine output < 250 mL/12 hours, no significant improvement (< 1 milligram per deciliter (mg/dL)) in serum creatinine from baseline value over the first 24 - 72 hours post-transplant, or dialysis treatment.
Time Frame: Randomization to Month 12
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants | 3.6 [1.2 to 6.1] | 0.4 [0.0 to 2.4] | 0.5 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Test type: Superiority or Other; Difference in Percent = -3.2, 95% CI 2-sided [-6.6 to -0.6] — For 95% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; Difference in Percent = -3.2, 95% CI 2-sided [-6.6 to -0.6] — For 95% CI of difference, normal approximation is used if N>=5 in both arms. Otherwise exact method is used

32. Secondary Outcome: Percent of Participants Using Lymphocyte Depleting Therapy (LDT) for the Initial Treatment of Acute Rejection (AR) by Month 36
Description: The use of LDT (thymoglobulin or antithymocyte gamma globulin [ATGAM]) was permitted only for participants randomized to cyclosporine (CsA) who experienced impaired renal allograft function and anticipated delayed graft function following transplantation. Acute rejection (AR) defined as a clinico-pathological event requiring clinical evidence (an unexplained rise of serum creatinine ≥ 25% from baseline creatinine or an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remained elevated within 14 days post-transplantation and clinical suspicion of acute rejection existed) and biopsy confirmation. AR defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Only the episode with the highest Banff grade for each participant was counted.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants
  Month 6 | 0.5 | 4.4 | 5.9
  Month 12 | 0.9 | 4.4 | 5.9
  Month 24 | 1.4 | 4.4 | 5.9
  Month 36 | 1.8 | 4.4 | 5.9

33. Secondary Outcome: Percent of Participants With Corticosteroid Resistant Acute Rejection (AR) by Month 36
Description: Steroid-resistant acute rejection (AR) defined as the use of lymphocyte-depletion therapy following treatment with corticosteroids. AR defined as a clinico-pathological event requiring clinical evidence and renal biopsy confirmation demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Clinical evidence defined: either a or b was satisfied: a) an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b) an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remained elevated within 14 days post-transplantation and clinical suspicion of acute rejection existed. Allograft biopsies were evaluated by a blinded central independent pathologist using Banff 97 international standardized histopathological working classification of kidney transplant pathology. Only the episode with the highest Banff grade for each participant was counted.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants
  Month 6 | 0.0 | 4.0 | 5.9
  Month 12 | 0.0 | 5.3 | 6.4
  Month 24 | 0.5 | 5.3 | 6.4
  Month 36 | 0.5 | 5.3 | 6.8

34. Secondary Outcome: Number of Participants Who Recovered Completely From an Episode of Acute Rejection (AR) by Month 12
Description: Acute rejection (AR) = a clinico-pathological event requiring clinical evidence and renal biopsy confirmation demonstrating a Banff 97 classification of Grade IA or greater. Clinical evidence = if either a or b was satisfied: a: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b: an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remains elevated within 14 days post-transplantation and clinical suspicion of acute rejection exists. Complete recovery following AR defined as serum creatinine [SCr] levels returned to baseline. Recovery calculated using 2 algorithms: Algorithm 1 = last laboratory measurement prior to onset of AR (baseline and first laboratory measurement after 84 days since onset of AR = resolution); Algorithm 2 = lowest laboratory measurement on or after transplantation and prior to onset day of AR (baseline and lowest laboratory measurement after onset on first AR up to Month 12 = resolution)
Time Frame: Randomization to Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with at least one episode of AR up to Month 12
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 16 | 39 | 48
participants
  Algorithm 1 | 13 | 29 | 39
  Algorithm 2 | 13 | 34 | 43

35. Secondary Outcome: Percent of Participants With Subclinical Rejection at Month 12
Description: Subclinical rejection defined as histological findings by the central pathologist consistent with acute rejection, but lacking its clinical correlate. Acute rejection defined as a clinico-pathological event requiring clinical evidence and renal biopsy confirmation demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection. Only the episode with the highest Banff grade for each participant was counted. Clinical evidence defined if either a or b was satisfied: a) an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; b) an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remained elevated within 14 days post-transplantation and clinical suspicion of acute rejection existed. Allograft biopsies were evaluated by a blinded central independent pathologist using Banff 97 working classification of kidney transplant pathology.
Time Frame: Month 12
Population: All randomized, transplanted, and treated participants; intent to treat (ITT) population with measurable component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 155 | 170 | 164
percentage of participants | 5.2 [1.7 to 8.6] | 4.7 [1.5 to 7.9] | 4.3 [1.2 to 7.4]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; Difference in Percent = -0.5, 97.3% CI 2-sided [-6.5 to 5.3]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Test type: Superiority or Other; Difference in Percent = -0.9, 97.3% CI 2-sided [-6.9 to 4.8]

36. Secondary Outcome: Number of Participants Treated for Acute Rejection (AR) Regardless of Histological Findings by Month 36
Description: Allograft rejection includes any episode of rejection including: clinically suspected rejection, treated rejection, any central biopsy-proven acute rejection (BPAR), and acute rejection (AR: a subset of BPAR) defined as central biopsy-proven rejection that was either clinically suspected by protocol-defined reasons or by other reasons and was treated. Acute rejection (AR) defined as a clinico-pathological event requiring clinical evidence ( either an unexplained rise of serum creatinine ≥ 25% from baseline creatinine or an unexplained decreased urine output; or fever and graft tenderness; or a serum creatinine that remained elevated within 14 days post-transplantation and clinical suspicion of AR) and renal biopsy confirmation biopsy demonstrating a Banff 97 working classification of kidney transplant pathology classification of Grade IA or greater, with higher scores indicating more severe rejection. Only the highest Banff grade for each participant was counted.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
participants
  Month 6 | 43 | 68 | 70
  Month 12 | 56 | 72 | 75
  Month 24 | 63 | 74 | 81
  Month 36 | 69 | 76 | 82

37. Secondary Outcome: Mean Value of Physical and Mental Components Using SF-36 Questionnaire
Description: SF-36 was a Participant-Reported Quality of Life (QoL) Short Form (SF) questionnaire measuring health-related quality of life (HRQL) covering 2 scale measures: physical component summary (PCS) and mental component summary (MCS). PCS represented by 4 domains: physical function, role limitations due to physical problems, pain, and general health perception. MCS represented by 4 domains: vitality, social function, role limitations due to emotional problems, and mental health. Their scores were computed based on weighted combinations of the 8 domain scores, which were transformed to a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Higher scores reflect better health-related functional status. Scoring is standardized using the norm-based scoring method where data is scored in relation to the U.S. general population having a mean of 50 and a standard deviation of 10. Scores below 50 are below the U.S. general population norm and above 50 are above the U.S. general population norm.
Time Frame: Months 6, 12, 24, 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 203 | 218 | 201
units on a scale
  Mental Component Score; Month 6 (n=191, 205, 189) | 49.4 (11.08) | 49.9 (10.55) | 51.1 (10.53)
  Physical Component Score; Month 6 (n=191,205,189) | 47.3 (8.91) | 48.9 (8.59) | 49.2 (7.58)
  Mental Component Score; Month 12 (n=198,210,194) | 49.5 (10.78) | 50.3 (10.08) | 49.9 (10.54)
  Physical Component Score; Month 12 (n=198,210,194) | 47.5 (9.34) | 49.6 (8.18) | 50.3 (8.21)
  Mental Component Score; Month 24 (n=200,214,198) | 48.3 (11.14) | 49.6 (10.77) | 48.8 (11.03)
  Physical Component Score; Month 24 (n=200,214,198) | 47.3 (9.50) | 49.0 (8.77) | 49.9 (8.03)
  Mental Component Score; Month 36 (n=203,218,201) | 46.9 (11.60) | 48.7 (11.26) | 48.3 (11.50)
  Physical Component Score; Month 36 (n=203,218,201) | 47.1 (9.47) | 49.2 (9.15) | 48.7 (8.90)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 6; Test type: Superiority or Other; p = 0.6573, ANOVA — Baseline observations were not used for imputations at subsequent time points; ANOVA model: Component Score = treatment. Missing values were imputed using last observation carried forward (LOCF) method; Mean Difference (Final Value) = 0.5, 95% CI 2-sided [-1.6 to 2.6] — Statistical tests comparing each belatacept regimen to the CsA regimen were conducted at a significance level of 0.05. Subjects with only baseline observations were excluded from these summaries
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 6; Test type: Superiority or Other; p = 0.1198, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.7, 95% CI 2-sided [-0.4 to 3.9] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 6; Test type: Superiority or Other; p = 0.0672, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.1 to 3.2] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 6; Test type: Superiority or Other; p = 0.0257, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [0.2 to 3.6] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 12; Test type: Superiority or Other; p = 0.4146, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.2 to 2.9] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 12; Test type: Superiority or Other; p = 0.7327, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 0.4, 95% CI 2-sided [-1.7 to 2.4] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 7: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 12; Test type: Superiority or Other; p = 0.0144, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 2.1, 95% CI 2-sided [0.4 to 3.8] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 8: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 12; Test type: Superiority or Other; p = 0.0015, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 2.8, 95% CI 2-sided [1.1 to 4.5] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 9: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 24; Test type: Superiority or Other; p = 0.2340, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.8 to 3.4] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 10: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 24; Test type: Superiority or Other; p = 0.6635, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 0.5, 95% CI 2-sided [-1.7 to 2.6] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 11: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 24; Test type: Superiority or Other; p = 0.0417, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.8, 95% CI 2-sided [0.1 to 3.5] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 12: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 24; Test type: Superiority or Other; p = 0.0026, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 2.7, 95% CI 2-sided [0.9 to 4.4] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 13: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 36; Test type: Superiority or Other; p = 0.0953, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.3 to 4.1] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 14: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 36; Test type: Superiority or Other; p = 0.1961, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.8 to 3.7] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 15: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 36; Test type: Superiority or Other; p = 0.0191, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 2.1, 95% CI 2-sided [0.3 to 3.9] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 16: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 36; Test type: Superiority or Other; p = 0.0684, ANOVA — Baseline observations were not used for imputations at subsequent time points; [statistical method as in outcome 37, analysis 1]; Mean Difference (Final Value) = 1.7, 95% CI 2-sided [-0.1 to 3.5] — [estimate comment as in outcome 37, analysis 1]

38. Secondary Outcome: Mean Value of the Eight Domain Scores of Quality of Life Using SF-36 Questionnaire
Description: as for outcome 37
Time Frame: Months 6, 12, 24, 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 205 | 219 | 206
units on a scale
  Bodily Pain, Month 6 (n=193, 207, 193) | 50.6 (10.96) | 52.5 (10.10) | 52.7 (10.04)
  General Health, Month 6 (n=193, 207, 194) | 47.9 (10.08) | 48.2 (9.67) | 49.0 (8.66)
  Mental Health, Month 6 (n=192, 206, 194) | 50.1 (11.08) | 50.3 (10.33) | 51.3 (10.78)
  Physical Functioning, Month 6 (n=193, 207, 194) | 47.4 (9.13) | 48.3 (9.01) | 48.0 (8.81)
  Role Emotional, Month 6 (n=192, 206, 191) | 44.6 (12.31) | 46.0 (11.19) | 46.8 (10.55)
  Role-Physical, Month 6 (n=192, 207, 192) | 43.2 (11.08) | 45.2 (10.34) | 46.7 (9.06)
  Social Functioning, Month 6 (n=193, 207, 194) | 47.5 (10.68) | 47.8 (10.41) | 47.9 (10.65)
  Vitality, Month 6 (n=192, 206, 194) | 54.0 (10.27) | 55.5 (9.75) | 56.2 (9.29)
  Bodily Pain, Month 12 (n=200, 213, 199) | 50.8 (10.79) | 52.7 (9.67) | 53.7 (9.60)
  General Health, Month 12 (n=200, 214, 199) | 46.9 (9.98) | 48.8 (9.57) | 49.2 (8.85)
  Mental Health, Month 12 (n=200, 213, 199) | 49.8 (10.99) | 50.7 (10.64) | 50.3 (10.29)
  Physical Functioning, Month 12 (n=200, 214, 198) | 47.2 (9.77) | 49.0 (8.88) | 48.1 (9.84)
  Role Emotional, Month 12 (n=198, 213, 196) | 45.8 (11.36) | 46.8 (10.82) | 45.9 (11.27)
  Role-Physical, Month 12 (n=199, 213, 196) | 45.0 (10.78) | 47.1 (10.00) | 47.5 (9.90)
  Social Functioning, Month 12 (n=200, 213, 199) | 47.6 (10.26) | 48.4 (9.61) | 49.1 (9.80)
  Vitality, Month 12 (n=200, 213, 199) | 53.3 (10.01) | 55.7 (9.81) | 56.0 (9.34)
  Bodily Pain, Month 24 (n=203, 219, 205) | 51.0 (10.82) | 51.4 (10.51) | 52.5 (10.47)
  General Health, Month 24 (n=203, 219, 205) | 46.2 (10.07) | 48.4 (9.61) | 48.7 (9.45)
  Mental Health, Month 24 (n=201, 215, 199) | 48.5 (11.13) | 49.7 (10.89) | 49.3 (10.85)
  Physical Functioning, Month 24 (n=203, 219, 205) | 46.5 (10.69) | 48.7 (9.76) | 48.0 (10.24)
  Role Emotional, Month 24 (n=202, 218, 205) | 44.8 (12.54) | 46.4 (10.89) | 46.0 (10.88)
  Role-Physical, Month 24 (n=203, 219, 204) | 44.1 (11.61) | 46.6 (10.39) | 48.0 (9.33)
  Social Functioning, Month 24 (n=203, 219, 205) | 47.3 (10.64) | 48.6 (10.28) | 47.7 (10.23)
  Vitality, Month 24 (n=201, 215, 200) | 52.5 (10.58) | 54.5 (10.30) | 54.2 (10.30)
  Bodily Pain, Month 36 (n=204, 219, 205) | 50.0 (11.40) | 52.3 (10.40) | 51.0 (11.05)
  General Health, Month 36 (n=205, 219, 206) | 45.5 (10.12) | 47.7 (10.45) | 47.5 (9.93)
  Mental Health, Month 36 (n=203, 219, 204) | 47.4 (11.64) | 48.9 (11.52) | 48.7 (11.43)
  Physical Functioning, Month 36 (n=204, 218, 206) | 46.8 (9.92) | 48.1 (10.22) | 47.8 (10.12)
  Role Emotional, Month 36 (n=204, 219, 205) | 43.5 (12.18) | 46.0 (11.85) | 45.3 (11.67)
  Role-Physical, Month 36 (n=204, 219, 205) | 43.6 (10.73) | 46.3 (11.03) | 46.2 (10.03)
  Social Functioning, Month 36 (n=204, 219, 206) | 46.6 (10.68) | 48.1 (10.28) | 47.1 (10.66)
  Vitality, Month 36 (n=203, 219, 204) | 51.4 (10.48) | 53.6 (11.38) | 53.4 (10.46)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Bodily Pain, Month 6; Test type: Superiority or Other; p = 0.0714, ANOVA; Domain Score = treatment; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.2 to 3.9] — Missing data were imputed by LOCF
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Bodily Pain, Month 6; Test type: Superiority or Other; p = 0.0536, ANOVA; Domain score = treatment; Mean Difference (Final Value) = 2.0, 95% CI 2-sided [-0.0 to 4.1] — Missing data were imputed by LOCF
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; General Health, Month 6; Test type: Superiority or Other; p = 0.7543, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.3, 95% CI 2-sided [-1.6 to 2.2] — Missing data were imputed by LOCF
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; General Health, Month 6; Test type: Superiority or Other; p = 0.2499, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.1, 95% CI 2-sided [-0.8 to 3.0] — Missing data were imputed by LOCF
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Mental Health, Month 6; Test type: Superiority or Other; p = 0.8332, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.2, 95% CI 2-sided [-1.9 to 2.3] — Missing data were imputed by LOCF
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Mental Health, Month 6; Test type: Superiority or Other; p = 0.2523, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.9 to 3.4] — Missing data were imputed by LOCF
Statistical Analysis 7: Comparison: Cyclosporine vs Belatacept LI; Physical Functioning, Month 6; Test type: Superiority or Other; p = 0.3018, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.9, 95% CI 2-sided [-0.8 to 2.7] — Missing data were imputed by LOCF
Statistical Analysis 8: Comparison: Cyclosporine vs Belatacept MI; Physical Functioning, Month 6; Test type: Superiority or Other; p = 0.5437, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.6, 95% CI 2-sided [-1.2 to 2.3] — Missing data were imputed by LOCF
Statistical Analysis 9: Comparison: Cyclosporine vs Belatacept LI; Role Emotional, Month 6; Test type: Superiority or Other; p = 0.2370, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.9 to 3.6] — Missing data were imputed by LOCF
Statistical Analysis 10: Comparison: Cyclosporine vs Belatacept MI; Role Emotional, Month 6; Test type: Superiority or Other; p = 0.0588, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [-0.1 to 4.5] — Missing data were imputed by LOCF
Statistical Analysis 11: Comparison: Cyclosporine vs Belatacept LI; Role Physical, Month 6; Test type: Superiority or Other; p = 0.0502, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.0, 95% CI 2-sided [-0.0 to 4.0] — Missing data were imputed by LOCF
Statistical Analysis 12: Comparison: Cyclosporine vs Belatacept MI; Role-Physical, Month 6; Test type: Superiority or Other; p = 0.0007, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 3.6, 95% CI 2-sided [1.5 to 5.6] — Missing data were imputed by LOCF
Statistical Analysis 13: Comparison: Cyclosporine vs Belatacept LI; Social Functioning, Month 6; Test type: Superiority or Other; p = 0.7637, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.3, 95% CI 2-sided [-1.8 to 2.4] — Missing data were imputed by LOCF
Statistical Analysis 14: Comparison: Cyclosporine vs Belatacept MI; Social Functioning, Month 6; Test type: Superiority or Other; p = 0.7006, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.4, 95% CI 2-sided [-1.7 to 2.5] — Missing data were imputed by LOCF
Statistical Analysis 15: Comparison: Cyclosporine vs Belatacept LI; Vitality, Month 6; Test type: Superiority or Other; p = 0.1222, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.4 to 3.4] — Missing data were imputed by LOCF
Statistical Analysis 16: Comparison: Cyclosporine vs Belatacept MI; Vitality, Month 6; Test type: Superiority or Other; p = 0.0289, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.2 to 4.1] — Missing data were imputed by LOCF
Statistical Analysis 17: Comparison: Cyclosporine vs Belatacept LI; Bodily Pain, Month 12; Test type: Superiority or Other; p = 0.0571, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.1 to 3.8] — Missing data were imputed by LOCF
Statistical Analysis 18: Comparison: Cyclosporine vs Belatacept MI; Bodily Pain, Month 12; Test type: Superiority or Other; p = 0.0042, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.9, 95% CI 2-sided [0.9 to 4.9] — Missing data were imputed by LOCF
Statistical Analysis 19: Comparison: Cyclosporine vs Belatacept LI; General Health, Month 12; Test type: Superiority or Other; p = 0.0423, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [0.1 to 3.7] — Missing data were imputed by LOCF
Statistical Analysis 20: Comparison: Cyclosporine vs Belatacept MI; General Health, Month 12; Test type: Superiority or Other; p = 0.0174, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.3, 95% CI 2-sided [0.4 to 4.1] — Missing data were imputed by LOCF
Statistical Analysis 21: Comparison: Cyclosporine vs Belatacept LI; Mental Health, Month 12; Test type: Superiority or Other; p = 0.3630, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.0, 95% CI 2-sided [-1.1 to 3.0] — Missing data were imputed by LOCF
Statistical Analysis 22: Comparison: Cyclosporine vs Belatacept MI; Mental Health, Month 12; Test type: Superiority or Other; p = 0.6319, ANOVA; Missing data were imputed by LOCF; Mean Difference (Final Value) = 0.5, 95% CI 2-sided [-1.6 to 2.6] — Missing data were imputed by LOCF
Statistical Analysis 23: Comparison: Cyclosporine vs Belatacept LI; Physical Functioning, Month 12; Test type: Superiority or Other; p = 0.0503, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.8, 95% CI 2-sided [-0.0 to 3.7] — Missing data were imputed by LOCF
Statistical Analysis 24: Comparison: Cyclosporine vs Belatacept MI; Physical Functioning, Month 12; Test type: Superiority or Other; p = 0.3291, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.9, 95% CI 2-sided [-0.9 to 2.8] — Missing data were imputed by LOCF
Statistical Analysis 25: Comparison: Cyclosporine vs Belatacept LI; Role Emotional, Month 12; Test type: Superiority or Other; p = 0.3860, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.0, 95% CI 2-sided [-1.2 to 3.1] — Missing data were imputed by LOCF
Statistical Analysis 26: Comparison: Cyclosporine vs Belatacept MI; Role Emotional, Month 12; Test type: Superiority or Other; p = 0.9672, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.0, 95% CI 2-sided [-2.2 to 2.3] — Missing data were imputed by LOCF
Statistical Analysis 27: Comparison: Cyclosporine vs Belatacept LI; Role-Physical, Month 12; Test type: Superiority or Other; p = 0.0392, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.1, 95% CI 2-sided [0.1 to 4.1] — Missing data were imputed by LOCF
Statistical Analysis 28: Comparison: Cyclosporine vs Belatacept MI; Role-Physical, Month 12; Test type: Superiority or Other; p = 0.0151, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.5, 95% CI 2-sided [0.5 to 4.5] — Missing data were imputed by LOCF
Statistical Analysis 29: Comparison: Cyclosporine vs Belatacept LI; Social Functioning, Month 12; Test type: Superiority or Other; p = 0.3978, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.1 to 2.7] — Missing data were imputed by LOCF
Statistical Analysis 30: Comparison: Cyclosporine vs Belatacept MI; Social Functioning, Month 12; Test type: Superiority or Other; p = 0.1263, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.4 to 3.5] — Missing data were imputed by LOCF
Statistical Analysis 31: Comparison: Cyclosporine vs Belatacept LI; Vitality, Month 12; Test type: Superiority or Other; p = 0.0160, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.3, 95% CI 2-sided [0.4 to 4.2] — Missing data were imputed by LOCF
Statistical Analysis 32: Comparison: Cyclosporine vs Belatacept MI; Vitality, Month 12; Test type: Superiority or Other; p = 0.0075, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.6, 95% CI 2-sided [0.7 to 4.5] — Missing data were imputed by LOCF
Statistical Analysis 33: Comparison: Cyclosporine vs Belatacept LI; Bodily Pain, Month 24; Test type: Superiority or Other; p = 0.6990, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.4, 95% CI 2-sided [-1.6 to 2.4] — Missing data were imputed by LOCF
Statistical Analysis 34: Comparison: Cyclosporine vs Belatacept MI; Bodily Pain, Month 24; Test type: Superiority or Other; p = 0.1608, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.6 to 3.5] — Missing data were imputed by LOCF
Statistical Analysis 35: Comparison: Cyclosporine vs Belatacept LI; General Health, Month 24; Test type: Superiority or Other; p = 0.0214, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.3 to 4.0] — Missing data were imputed by LOCF
Statistical Analysis 36: Comparison: Cyclosporine vs Belatacept MI; General Health, Month 24; Test type: Superiority or Other; p = 0.00886, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.5, 95% CI 2-sided [0.6 to 4.4] — Missing data were imputed by LOCF
Statistical Analysis 37: Comparison: Cyclosporine vs Belatacept LI; Mental Health, Month 24; Test type: Superiority or Other; p = 0.2555, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.2, 95% CI 2-sided [-0.9 to 3.3] — Missing data were imputed by LOCF
Statistical Analysis 38: Comparison: Cyclosporine vs Belatacept MI; Mental Health, Month 24; Test type: Superiority or Other; p = 0.4804, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.4 to 2.9] — Missing data were imputed by LOCF
Statistical Analysis 39: Comparison: Cyclosporine vs Belatacept LI; Physical Functioning, Month 24; Test type: Superiority or Other; p = 0.0276, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.2 to 4.2] — Missing data were imputed by LOCF
Statistical Analysis 40: Comparison: Cyclosporine vs Belatacept MI; Physical Functioning, Month 24; Test type: Superiority or Other; p = 0.1285, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.4 to 3.5] — Missing data were imputed by LOCF
Statistical Analysis 41: Comparison: Cyclosporine vs Belatacept LI; Role Emotional, Month 24; Test type: Superiority or Other; p = 0.1352, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.7, 95% CI 2-sided [-0.5 to 3.9] — Missing data were imputed by LOCF
Statistical Analysis 42: Comparison: Cyclosporine vs Belatacept MI; Role Emotional, Month 24; Test type: Superiority or Other; p = 0.2663, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-1.0 to 3.5] — Missing data were imputed by LOCF
Statistical Analysis 43: Comparison: Cyclosporine vs Belatacept LI; Role-Physical, Month 24; Test type: Superiority or Other; p = 0.0164, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.5, 95% CI 2-sided [0.5 to 4.5] — Missing data were imputed by LOCF
Statistical Analysis 44: Comparison: Cyclosporine vs Belatacept MI; Role-Physical, Month 24; Test type: Superiority or Other; p = 0.0002, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 3.9, 95% CI 2-sided [1.9 to 5.9] — Missing data were imputed by LOCF
Statistical Analysis 45: Comparison: Cyclosporine vs Belatacept LI; Social Functioning, Month 24; Test type: Superiority or Other; p = 0.1914, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.7 to 3.3] — Missing data were imputed by LOCF
Statistical Analysis 46: Comparison: Cyclosporine vs Belatacept MI; Social Functioning, Month 24; Test type: Superiority or Other; p = 0.6882, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.4, 95% CI 2-sided [-1.6 to 2.4] — Missing data were imputed by LOCF
Statistical Analysis 47: Comparison: Cyclosporine vs Belatacept LI; Vitality, Month 24; Test type: Superiority or Other; p = 0.0547, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.0, 95% CI 2-sided [-0.0 to 4.0] — Missing data were imputed by LOCF
Statistical Analysis 48: Comparison: Cyclosporine vs Belatacept MI; Vitality, Month 24; Test type: Superiority or Other; p = 0.0992, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.7, 95% CI 2-sided [-0.3 to 3.8] — Missing data were imputed by LOCF
Statistical Analysis 49: Comparison: Cyclosporine vs Belatacept LI; Bodily Pain, Month 36; Test type: Superiority or Other; p = 0.0339, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.3, 95% CI 2-sided [0.2 to 4.4] — Missing data were imputed by LOCF
Statistical Analysis 50: Comparison: Cyclosporine vs Belatacept MI; Bodily Pain, Month 36; Test type: Superiority or Other; p = 0.3572, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.0, 95% CI 2-sided [-1.1 to 3.1] — Missing data were imputed by LOCF
Statistical Analysis 51: Comparison: Cyclosporine vs Belatacept LI; General Health, Month 36; Test type: Superiority or Other; p = 0.0211, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.3, 95% CI 2-sided [0.3 to 4.2] — Missing data were imputed by LOCF
Statistical Analysis 52: Comparison: Cyclosporine vs Belatacept MI; General Health, Month 36; Test type: Superiority or Other; p = 0.0450, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.0, 95% CI 2-sided [0.0 to 4.0] — Missing data were imputed by LOCF
Statistical Analysis 53: Comparison: Cyclosporine vs Belatacept LI; Mental Health, Month 36; Test type: Superiority or Other; p = 0.1710, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.7 to 3.7] — Missing data were imputed by LOCF
Statistical Analysis 54: Comparison: Cyclosporine vs Belatacept MI; Mental Health, Month 36; Test type: Superiority or Other; p = 0.2484, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.9 to 3.6] — Missing data were imputed by LOCF
Statistical Analysis 55: Comparison: Cyclosporine vs Belatacept LI; Physical Functioning, Month 36; Test type: Superiority or Other; p = 0.1836, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.6 to 3.2] — Missing data were imputed by LOCF
Statistical Analysis 56: Comparison: Cyclosporine vs Belatacept MI; Physical Functioning, Month 36; Test type: Superiority or Other; p = 0.3303, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.0, 95% CI 2-sided [-1.0 to 2.9] — Missing data were imputed by LOCF
Statistical Analysis 57: Comparison: Cyclosporine vs Belatacept LI; Role Emotional, Month 36; Test type: Superiority or Other; p = 0.0299, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.5, 95% CI 2-sided [0.2 to 4.8] — Missing data were imputed by LOCF
Statistical Analysis 58: Comparison: Cyclosporine vs Belatacept MI; Role Emotional, Month 36; Test type: Superiority or Other; p = 0.1141, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.4 to 4.2] — Missing data were imputed by LOCF
Statistical Analysis 59: Comparison: Cyclosporine vs Belatacept LI; Role-Physical, Month 36; Test type: Superiority or Other; p = 0.0087, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.7, 95% CI 2-sided [0.7 to 4.7] — Missing data were imputed by LOCF
Statistical Analysis 60: Comparison: Cyclosporine vs Belatacept MI; Role-Physical, Month 36; Test type: Superiority or Other; p = 0.0128, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.6, 95% CI 2-sided [0.6 to 4.7] — Missing data were imputed by LOCF
Statistical Analysis 61: Comparison: Cyclosporine vs Belatacept LI; Social Functioning, Month 36; Test type: Superiority or Other; p = 0.1369, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 1.5, 95% CI 2-sided [-0.5 to 3.5] — Missing data were imputed by LOCF
Statistical Analysis 62: Comparison: Cyclosporine vs Belatacept MI; Social Functioning, Month 36; Test type: Superiority or Other; p = 0.6331, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 0.5, 95% CI 2-sided [-1.5 to 2.5] — Missing data were imputed by LOCF
Statistical Analysis 63: Comparison: Cyclosporine vs Belatacept LI; Vitality, Month 36; Test type: Superiority or Other; p = 0.0361, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.1 to 4.3] — Missing data were imputed by LOCF
Statistical Analysis 64: Comparison: Cyclosporine vs Belatacept MI; Vitality, Month 36; Test type: Superiority or Other; p = 0.0525, ANOVA; Missing data = treatment; Mean Difference (Final Value) = 2.1, 95% CI 2-sided [-0.0 to 4.2] — Missing data were imputed by LOCF

39. Secondary Outcome: Mean Relative to an Identified Distribution (Ridit) Value of Symptom Occurrence and Symptom Distress Using Modified Transplant Symptom Occurrence and Symptom Distress Scale (MTSOSDS-59R)
Description: The Modified Transplant Symptom Occurrence and Symptom Distress Scale (MTSOSD-59R) was used to assess the occurrence (never, occasionally, regularly, almost always, always) and distress (0=no distress to 4=terrible distress) of symptoms associated with immunosuppressive therapies. Ridit (relative to an identified distribution) analysis (Fleiss JL. Statistical methods for rates and proportions. New York: John Wiley & Sons, Inc. 1991) was used. Ridit scores were calculated at baseline and at 6, 12, 24, and 36 months for overall symptom occurrence score and overall symptom distress. The Ridit score reflects the probability that a score observed for an individual randomly selected from a group would be higher (worse symptom) than a score observed for a randomly selected individual from the reference group. The reference group was constituted by the frequency distribution of the responses of all participants on all items at baseline. The ridit of the reference group is by definition, 0.5.
Time Frame: Months 6, 12, 24, 36
Population: All randomized and transplanted participants, intent to treat (ITT) population.
Measure: Mean (Standard Error); unit: Ridit score
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 186 | 197 | 187
Ridit score
  Symptom Distress, Month 6 (n=157, 164, 155) | 0.4643 (0.00452) | 0.4407 (0.00404) | 0.4451 (0.00422)
  Symptom Occurrence, Month 6 (n=166, 176, 165) | 0.4721 (0.00463) | 0.4495 (0.00425) | 0.4459 (0.00432)
  Symptom Distress, Month 12 (n=169, 185, 169) | 0.4751 (0.00453) | 0.4510 (0.00397) | 0.4546 (0.00421)
  Symptom Occurrence, Month 12 (n=173, 188, 173) | 0.4776 (0.00458) | 0.4519 (0.00411) | 0.4525 (0.00430)
  Symptom Distress, Month 24 (n=182, 195, 179) | 0.4798 (0.00443) | 0.4584 (0.00397) | 0.4646 (0.00424)
  Symptom Occurrence, Month 24 (n=184, 197, 184) | 0.4804 (0.00446) | 0.4574 (0.00406) | 0.4593 (0.00423)
  Symptom Distress, Month 36 (n=184, 196, 183) | 0.5000 (0.00456) | 0.4746 (0.00408) | 0.4892 (0.00442)
  Symptom Occurrence, Month 36 (n=186, 197, 187) | 0.5000 (0.00459) | 0.4732 (0.00421) | 0.4846 (0.00441)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Symptom Distress, Month 6. For calculation of symptom distress, those symptoms that never occurred will be converted to missing values, in order to avoid anticipatory symptom distress; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.024, 95% CI 2-sided [-0.032 to -0.015]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; [analysis description as in outcome 39, analysis 1]; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.019, 95% CI 2-sided [-0.028 to -0.011]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Symptom Occurrence, Month 6; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.023, 95% CI 2-sided [-0.031 to -0.014]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Symptom Occurrence, Month 6; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.026, 95% CI 2-sided [-0.035 to -0.017]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Symptom Distress, Month 12. For calculation of symptom distress, those symptoms that never occurred will be converted to missing values, in order to avoid anticipatory symptom distress; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.024, 95% CI 2-sided [-0.032 to -0.016]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; [analysis description as in outcome 39, analysis 5]; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.020, 95% CI 2-sided [-0.029 to -0.012]
Statistical Analysis 7: Comparison: Cyclosporine vs Belatacept LI; Symptom Occurrence, Month 12; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.026, 95% CI 2-sided [-0.034 to -0.017]
Statistical Analysis 8: Comparison: Cyclosporine vs Belatacept MI; Symptom Occurrence, Month 12; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.025, 95% CI 2-sided [-0.034 to -0.016]
Statistical Analysis 9: Comparison: Cyclosporine vs Belatacept LI; Symptom Distress, Month 24. For calculation of symptom distress, those symptoms that never occurred will be converted to missing values, in order to avoid anticipatory symptom distress; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.021, 95% CI 2-sided [-0.030 to -0.013]
Statistical Analysis 10: Comparison: Cyclosporine vs Belatacept MI; [analysis description as in outcome 39, analysis 9]; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.015, 95% CI 2-sided [-0.024 to -0.007]
Statistical Analysis 11: Comparison: Cyclosporine vs Belatacept LI; Symptom Occurrence, Month 24; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.023, 95% CI 2-sided [-0.031 to -0.015]
Statistical Analysis 12: Comparison: Cyclosporine vs Belatacept MI; Symptom Occurrence, Month 24; Test type: Superiority or Other; p < 0.0001, z-test — Missing data were imputed by LOCF. The ridit of the reference group is by definition 0.5; The obtained ridits between treatment groups will be compared using z-test at 0.05 significance level for each year; Mean Difference (Final Value) = -0.021, 95% CI 2-sided [-0.030 to -0.013]

40. Secondary Outcome: Mean Changes in the Value of Physical and Mental Components Using SF-36 From Baseline Up To Months 6, 12, 24, and 36
Description: as for outcome 37
Time Frame: Baseline to Months 6, 12, 24,and 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 192 | 203 | 193
units on a scale
  Mental Component Score; Month 6 (n=187, 197, 184) | 5.4 (0.714) | 6.2 (0.695) | 7.3 (0.720)
  Physical Component Score; Month 6 (n=187, 197, 184 | 5.0 (0.580) | 6.2 (0.566) | 6.7 (0.585)
  Mental Component Score; Month 12 (n=192, 200, 189) | 5.4 (0.687) | 6.8 (0.673) | 6.2 (0.693)
  Physical Component Score; Month 12 (n=192,200,189) | 5.5 (0.589) | 7.1 (0.577) | 7.8 (0.594)
  Mental Component Score; Month 24 (n=191,202,193) | 4.4 (0.732) | 5.7 (0.712) | 5.1 (0.728)
  Physical Component Score; Month 24 (n=191,202,193) | 5.1 (0.601) | 6.5 (0.584) | 7.3 (0.597)
  Mental Component Score; Month 36 (n=190,203,191) | 2.6 (0.756) | 5.1 (0.732) | 4.5 (0.754)
  Physical Component Score; Month 36 (n=190,203,191) | 4.9 (0.633) | 6.5 (0.612) | 6.1 (0.631)
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 6; Test type: Superiority or Other; p = 0.4498, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.2 to 2.7] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 6; Test type: Superiority or Other; p = 0.0584, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.1 to 3.9] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 6; Test type: Superiority or Other; p = 0.1595, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.1, 95% CI 2-sided [-0.5 to 2.7] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 6; Test type: Superiority or Other; p = 0.0457, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.7, 95% CI 2-sided [0.0 to 3.3] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 12; Test type: Superiority or Other; p = 0.1729, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.3, 95% CI 2-sided [-0.6 to 3.2] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 12; Test type: Superiority or Other; p = 0.4209, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.1 to 2.7] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 7: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 12; Test type: Superiority or Other; p = 0.0526, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.6, 95% CI 2-sided [-0.0 to 3.2] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 8: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 12; Test type: Superiority or Other; p = 0.0077, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.6 to 3.9] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 9: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 24; Test type: Superiority or Other; p = 0.1849, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.4, 95% CI 2-sided [-0.6 to 3.4] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 10: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 24; Test type: Superiority or Other; p = 0.4633, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 0.8, 95% CI 2-sided [-1.3 to 2.8] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 11: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 24; Test type: Superiority or Other; p = 0.0971, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.4, 95% CI 2-sided [-0.3 to 3.0] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 12: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 24; Test type: Superiority or Other; p = 0.0102, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 2.2, 95% CI 2-sided [0.5 to 3.8] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 13: Comparison: Cyclosporine vs Belatacept LI; Mental Component Score; Month 36; Test type: Superiority or Other; p = 0.0186, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 2.5, 95% CI 2-sided [0.4 to 4.5] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 14: Comparison: Cyclosporine vs Belatacept MI; Mental Component Score; Month 36; Test type: Superiority or Other; p = 0.0775, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.9, 95% CI 2-sided [-0.2 to 4.0] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 15: Comparison: Cyclosporine vs Belatacept LI; Physical Component Score; Month 36; Test type: Superiority or Other; p = 0.0768, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.6, 95% CI 2-sided [-0.2 to 3.3] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 16: Comparison: Cyclosporine vs Belatacept MI; Physical Component Score; Month 36; Test type: Superiority or Other; p = 0.1876, ANCOVA; Adjusted mean based on an ANCOVA model with treatment as factor, and baseline value as covariate; Mean Difference (Final Value) = 1.2, 95% CI 2-sided [-0.6 to 2.9] — [estimate comment as in outcome 37, analysis 1]

41. Secondary Outcome: Mean Change in the Value of the Eight Domain Scores Using SF-36 From Baseline Up To Months 6, 12, 24, and 36
Description: as for outcome 37
Time Frame: Baseline to Months 6, 12, 24, and 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 194 | 207 | 197
units on a scale
  Bodily Pain, Month 6 (n=189,201,189) | 2.9 (0.712) | 4.5 (0.691) | 4.6 (0.712)
  General Health, Month 6 (n=189,201,190) | 6.7 (0.631) | 7.1 (0.612) | 7.3 (0.630)
  Mental Health, Month 6 (n=188,198,190) | 4.7 (0.716) | 5.2 (0.698) | 6.1 (0.712)
  Physical Functioning, Month 6 (n=189,201,190) | 4.7 (0.610) | 5.3 (0.592) | 5.6 (0.610)
  Role Emotional, Month 6 (n=188,200,186) | 4.7 (0.767) | 5.8 (0.744) | 6.9 (0.772)
  Role-Physical, Month 6 (n=188,201,187) | 6.4 (0.718) | 8.4 (0.694) | 9.6 (0.720)
  Social Functioning, Month 6 (n=189,201,190) | 6.0 (0.724) | 6.8 (0.702) | 6.9 (0.722)
  Vitality, Month 6 (n=188,198,190) | 7.5 (0.668) | 9.0 (0.651) | 9.9 (0.665)
  Bodily Pain, Month 12 (n=194,205,195) | 3.1 (0.665) | 4.8 (0.647) | 5.5 (0.664)
  General Health, Month 12 (n=194,206,195) | 6.0 (0.638) | 7.7 (0.619) | 7.6 (0.636)
  Mental Health, Month 12 (n=194,203,195) | 4.4 (0.685) | 6.0 (0.670) | 5.0 (0.684)
  Physical Functioning, Month 12 (n=194,206,194) | 4.7 (0.640) | 6.2 (0.621) | 5.8 (0.641)
  Role Emotional, Month 12 (n=192,205,191) | 5.7 (0.765) | 6.6 (0.741) | 5.9 (0.768)
  Role-Physical, Month 12 (n=193,205,191) | 8.3 (0.716) | 10.3 (0.695) | 10.4 (0.720)
  Social Functioning, Month 12 (n=194,205,195) | 6.4 (0.669) | 7.7 (0.650) | 8.0 (0.667)
  Vitality, Month 12 (n=194,203,195) | 7.0 (0.651) | 9.2 (0.636) | 9.7 (0.649)
  Bodily Pain, Month 24 (n=192,207,197) | 3.2 (0.722) | 3.3 (0.696) | 4.1 (0.713)
  General Health, Month 24 (n=193,207,197) | 5.1 (0.641) | 7.2 (0.619) | 6.8 (0.635)
  Mental Health, Month 24 (n=193,203,195) | 3.2 (0.710) | 4.6 (0.692) | 4.0 (0.706)
  Physical Functioning, Month 24 (n=193,207,197) | 4.1 (0.685) | 5.7 (0.662) | 5.5 (0.679)
  Role Emotional, Month 24 (n=192,206,196) | 4.7 (0.793) | 6.0 (0.766) | 5.9 (0.785)
  Role-Physical, Month 24 (n=193,207,195) | 7.4 (0.740) | 9.4 (0.715) | 10.7 (0.737)
  Social Functioning, Month 24 (n=193, 207,197) | 5.9 (0.722) | 7.4 (0.697) | 6.3 (0.715)
  Vitality, Month 24 (n=193,203,196) | 6.2 (0.700) | 7.9 (0.682) | 8.0 (0.695)
  Bodily Pain, Month 36 (n=191,207,196) | 2.3 (0.739) | 4.2 (0.710) | 3.0 (0.730)
  General Health, Month 36 (n=193,207,197) | 4.1 (0.681) | 6.6 (0.657) | 5.8 (0.674)
  Mental Health, Month 36 (n=191,204,195) | 1.8 (0.754) | 4.1 (0.729) | 3.4 (0.746)
  Physical Functioning, Month 36 (n=192,206,197) | 4.4 (0.692) | 5.3 (0.668) | 5.1 (0.684)
  Role Emotional, Month 36 (n=192,207,195) | 3.3 (0.830) | 5.6 (0.800) | 5.0 (0.824)
  Role-Physical, Month 36 (n=192,207,195) | 6.8 (0.754) | 9.2 (0.727) | 8.9 (0.749)
  Social Functioning, Month 36 (n=192,207,197) | 5.1 (0.736) | 7.0 (0.708) | 5.6 (0.726)
  Vitality, Month 36 (n=191,204,195) | 4.9 (0.721) | 7.3 (0.698) | 7.3 (0.714)

42. Secondary Outcome: Percent of Participants Surviving With a Functioning Graft
Description: Graft loss was defined as either functional loss or physical loss (nephrectomy). Functional loss was defined as a sustained level of serum creatinine (SCr) ≥ 6.0 milligrams per deciliter (mg/dL) or 530 micromoles per liter (μmol/L) as determined by the central laboratory for ≥ 4 weeks or ≥ 56 consecutive days of dialysis or impairment of renal function to such a degree that the participant underwent retransplant.
Time Frame: Months 24, 36
Population: All randomized and transplanted participants, intent to treat (ITT) population. For 95% CI within each group, normal approximation is used in N>=5. Otherwise exact method is used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants
  Month 24 | 90.5 [86.6 to 94.4] | 94.7 [91.8 to 97.6] | 94.1 [90.9 to 97.2]
  Month 36 | 88.7 [84.5 to 92.9] | 92.0 [88.5 to 95.6] | 92.2 [88.7 to 95.8]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 24; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Percent = 4.2, 97.3% CI 2-sided [-1.3 to 10.1]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 24; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Percent = 3.6, 97.3% CI 2-sided [-2.2 to 9.6]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Month 36; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Percent = 3.3, 97.3% CI 2-sided [-2.9 to 9.8]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in Percent = 3.5, 97.3% CI 2-sided [-2.8 to 10.0]

43. Secondary Outcome: Percent of Participants With Composite Endpoint or Death, Graft Loss or Acute Rejection by Month 36
Description: Graft loss was defined as either functional loss or physical loss (nephrectomy). Functional loss was defined as a sustained level of serum creatinine (SCr) ≥ 6.0 milligrams per deciliter (mg/dL) or 530 micromoles per liter (μmol/L) as determined by the central laboratory for ≥ 4 weeks or ≥ 56 consecutive days of dialysis or impairment of renal function to such a degree that the participant underwent retransplant. Acute rejection was defined as central biopsy proven rejection that was either (1) clinically suspected by protocol defined reasons or (2) clinically suspected by other reasons and treated. Death and graft loss were not imputed.
Time Frame: Randomization to Month 36
Population: All randomized and transplanted participants, intent to treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclosporine | Belatacept LI | Belatacept MI
Number analyzed (Participants) | 221 | 226 | 219
percentage of participants
  Month 12 | 13.6 [9.1 to 18.1] | 19.5 [14.3 to 24.6] | 25.1 [19.4 to 30.9]
  Month 24 | 18.1 [13.0 to 23.2] | 19.9 [14.7 to 25.1] | 27.9 [21.9 to 33.8]
  Month 36 | 19.9 [14.6 to 25.2] | 20.8 [15.5 to 26.1] | 28.3 [22.3 to 34.3]
Statistical Analysis 1: Comparison: Cyclosporine vs Belatacept LI; Month 12; Test type: Superiority or Other; Difference in Percent = 5.9, 95% CI 2-sided [-1.0 to 12.8]
Statistical Analysis 2: Comparison: Cyclosporine vs Belatacept MI; Month 12; Test type: Superiority or Other; Difference in Percent = 11.5, 95% CI 2-sided [4.2 to 18.9]
Statistical Analysis 3: Comparison: Cyclosporine vs Belatacept LI; Month 24; Test type: Superiority or Other; Difference in Percent = 1.8, 95% CI 2-sided [-5.5 to 9.1]
Statistical Analysis 4: Comparison: Cyclosporine vs Belatacept MI; Month 24; Test type: Superiority or Other; Difference in Percent = 9.8, 95% CI 2-sided [1.9 to 17.6]
Statistical Analysis 5: Comparison: Cyclosporine vs Belatacept LI; Month 36; Test type: Superiority or Other; Difference in Percent = 0.9, 95% CI 2-sided [-6.6 to 8.4]
Statistical Analysis 6: Comparison: Cyclosporine vs Belatacept MI; Month 36; Test type: Superiority or Other; Difference in Percent = 8.4, 95% CI 2-sided [0.4 to 16.4]

ADVERSE EVENTS:
Time Frame: Randomization to Long Term Extension, up to 84 Months
Description: Study start: March 2005; Study Completion: April 2015. All randomized, transplanted, and treated participants (ITT population)
Groups:
- Belatacept - LI: Belatacept LI (less intensive): solution, intravenous (IV), 10 milligrams/kilogram (mg/kg): Days 1 and 5, Weeks 2, 4, 8 and 12, then 5 mg/kg every (q) 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
- Belatacept - MI: Belatacept MI (more intensive): solution, IV, 10mg/kg: Days 1 and 5, Weeks 2, 4, 6, 8, 10,12, 16, 20, and 24, then 5 milligrams/kilogram (mg/kg) every 4 weeks, q 4 weeks, 36 months (ST), 5 mg/kg every 4 weeks, q 4 weeks, 24 months (LT)
Arm/Group | Cyclosporine | Belatacept - LI | Belatacept - MI
Serious Adverse Events (participants affected / at risk) | 167/215 | 160/226 | 164/219
Other Adverse Events (participants affected / at risk) | 213/215 | 222/226 | 216/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=215) | Belatacept - LI (N=226) | Belatacept - MI (N=219)
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Acinetobacter infection (Infections and infestations) | 0 | 1 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 13 | 4 | 6
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 1 | 1
Arteriovenous graft site infection (Infections and infestations) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 3
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Blood glucose fluctuation (Investigations) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 5 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Delayed graft function (Injury, poisoning and procedural complications) | 9 | 3 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Encephalitis meningococcal (Infections and infestations) | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 2
Furuncle (Infections and infestations) | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 2 | 2 | 2
Headache (Nervous system disorders) | 2 | 1 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 2
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 2 | 3
Hyperthermia (General disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Infarction (Vascular disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 4
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Pneumatosis (General disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 4 | 6
Renal artery thrombosis (Renal and urinary disorders) | 0 | 0 | 2
Renal lymphocele (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Transplant dysfunction (Injury, poisoning and procedural complications) | 7 | 5 | 3
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 3
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 2
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3
Vulval abscess (Infections and infestations) | 0 | 0 | 1
Accidental death (General disorders) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 2
Cellulitis (Infections and infestations) | 4 | 4 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 7 | 4 | 9
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 5
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 3
Hernia (General disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Iris neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphocele (Vascular disorders) | 8 | 2 | 2
Meningitis cryptococcal (Infections and infestations) | 0 | 1 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 7 | 4
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 1 | 2
Renal impairment (Renal and urinary disorders) | 6 | 7 | 5
Renal transplant failure (Immune system disorders) | 0 | 2 | 0
Renal tubular disorder (Renal and urinary disorders) | 2 | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 3
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal urinary tract infection (Infections and infestations) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site infection (Infections and infestations) | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 9 | 8
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Blastomycosis (Infections and infestations) | 0 | 0 | 1
Blood creatine increased (Investigations) | 1 | 2 | 1
Blood culture positive (Investigations) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 2 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Embolism venous (Vascular disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 5 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Osteomyelitis (Infections and infestations) | 1 | 1 | 2
Ovarian abscess (Infections and infestations) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral artery dissection (Vascular disorders) | 1 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 2 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Polycystic liver disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Polyomavirus test positive (Investigations) | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sepsis (Infections and infestations) | 8 | 6 | 9
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 5 | 2 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Vascular compression (Vascular disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0
West Nile viral infection (Infections and infestations) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 3 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 8 | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 2 | 5
Diabetic foot infection (Infections and infestations) | 0 | 1 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 3 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Malaria (Infections and infestations) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 0 | 1
Papilloedema (Eye disorders) | 1 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 3 | 2
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Renal artery stenosis (Renal and urinary disorders) | 2 | 2 | 3
Renal mass (Renal and urinary disorders) | 2 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 4 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0
Septic shock (Infections and infestations) | 3 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 4
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 2 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 4 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 3 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abscess (Infections and infestations) | 2 | 0 | 0
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 7
Appendicitis (Infections and infestations) | 1 | 1 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 12 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 4 | 0 | 4
Incarcerated hernia (General disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 1 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 2 | 2
Pneumocystis test positive (Investigations) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 16 | 17 | 13
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 3 | 3 | 2
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8 | 9
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Thymic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Ultrasound kidney abnormal (Investigations) | 1 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 4 | 2
Wound evisceration (Injury, poisoning and procedural complications) | 2 | 2 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 5
Chest discomfort (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cryptococcosis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 2
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 1 | 2
Hepatic cyst infection (Infections and infestations) | 0 | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 2 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Influenza (Infections and infestations) | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pineal gland cyst (Nervous system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 17 | 14 | 9
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Splenic cyst (Blood and lymphatic system disorders) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Strongyloidiasis (Infections and infestations) | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 3 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1 | 0
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 1 | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 32 | 26 | 21
Urinary tract infection bacterial (Infections and infestations) | 3 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Action tremor (Nervous system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 5 | 6
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chest pain (General disorders) | 6 | 3 | 6
Coagulation test abnormal (Investigations) | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 3 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 4 | 2 | 5
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 3
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parasitic encephalitis (Infections and infestations) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 3 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 9 | 9 | 8
Pyelonephritis viral (Infections and infestations) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular atrophy (Renal and urinary disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Urinary fistula (Renal and urinary disorders) | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1 | 0
Urinoma (Renal and urinary disorders) | 2 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 1 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0
BK virus infection (Infections and infestations) | 1 | 1 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 1 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 16 | 10 | 5
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0 | 0
Chronic allograft nephropathy (Immune system disorders) | 4 | 4 | 4
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Cytomegalovirus duodenitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus enteritis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 8 | 13 | 16
Device related infection (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 1 | 0
Graft loss (Injury, poisoning and procedural complications) | 2 | 4 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 2 | 1 | 0
Infection (Infections and infestations) | 0 | 2 | 2
Influenza like illness (General disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Ischaemic ulcer (General disorders) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0
Mononeuropathy (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 2 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Orchitis (Infections and infestations) | 1 | 1 | 1
Pertussis (Infections and infestations) | 0 | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 9 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 1
Ureteral necrosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 4 | 2 | 3
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=215) | Belatacept - LI (N=226) | Belatacept - MI (N=219)
Delayed graft function (Injury, poisoning and procedural complications) | 28 | 26 | 22
Dysuria (Renal and urinary disorders) | 34 | 26 | 34
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 19 | 11
Haematoma (Vascular disorders) | 16 | 9 | 12
Headache (Nervous system disorders) | 46 | 75 | 65
Hyperkalaemia (Metabolism and nutrition disorders) | 44 | 41 | 18
Hypertension (Vascular disorders) | 82 | 87 | 70
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11 | 6 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 25 | 27 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 15 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 49 | 48
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 7 | 6
Leukopenia (Blood and lymphatic system disorders) | 37 | 48 | 40
Metabolic acidosis (Metabolism and nutrition disorders) | 19 | 8 | 13
Nausea (Gastrointestinal disorders) | 70 | 62 | 59
Oedema (General disorders) | 25 | 11 | 13
Transplant dysfunction (Injury, poisoning and procedural complications) | 12 | 7 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 9 | 21 | 17
Vomiting (Gastrointestinal disorders) | 46 | 55 | 45
Chills (General disorders) | 10 | 15 | 9
Contusion (Injury, poisoning and procedural complications) | 8 | 8 | 11
Dizziness (Nervous system disorders) | 32 | 25 | 24
Fall (Injury, poisoning and procedural complications) | 16 | 11 | 10
Fungal skin infection (Infections and infestations) | 9 | 16 | 10
Gastroenteritis (Infections and infestations) | 20 | 19 | 25
Haematuria (Renal and urinary disorders) | 41 | 39 | 33
Hypoaesthesia (Nervous system disorders) | 7 | 19 | 12
Leukocyturia (Renal and urinary disorders) | 9 | 13 | 6
Oedema peripheral (General disorders) | 87 | 70 | 64
Pain (General disorders) | 14 | 14 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 40 | 36
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 10
Renal impairment (Renal and urinary disorders) | 14 | 10 | 7
Skin lesion (Skin and subcutaneous tissue disorders) | 15 | 22 | 24
Tinnitus (Ear and labyrinth disorders) | 7 | 12 | 5
Weight increased (Investigations) | 24 | 24 | 27
Bradycardia (Cardiac disorders) | 13 | 9 | 8
Conjunctivitis (Infections and infestations) | 9 | 11 | 12
Depression (Psychiatric disorders) | 18 | 17 | 26
Flatulence (Gastrointestinal disorders) | 11 | 16 | 9
Gingival hyperplasia (Gastrointestinal disorders) | 18 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 | 31 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 42 | 38 | 42
Hypomagnesaemia (Metabolism and nutrition disorders) | 24 | 17 | 18
Incision site pain (Injury, poisoning and procedural complications) | 38 | 30 | 33
Insomnia (Psychiatric disorders) | 38 | 39 | 42
Onychomycosis (Infections and infestations) | 10 | 16 | 15
Oral herpes (Infections and infestations) | 12 | 22 | 16
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 9 | 14
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 9 | 14
Tachycardia (Cardiac disorders) | 23 | 12 | 19
Abdominal discomfort (Gastrointestinal disorders) | 11 | 7 | 8
Abdominal pain upper (Gastrointestinal disorders) | 24 | 22 | 19
Acne (Skin and subcutaneous tissue disorders) | 31 | 22 | 23
Bronchitis (Infections and infestations) | 21 | 29 | 22
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 13 | 10 | 7
Constipation (Gastrointestinal disorders) | 68 | 83 | 65
Dehydration (Metabolism and nutrition disorders) | 15 | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 26 | 35 | 20
Herpes zoster (Infections and infestations) | 19 | 14 | 20
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 | 15 | 8
Paraesthesia (Nervous system disorders) | 19 | 18 | 7
Polycythaemia (Blood and lymphatic system disorders) | 11 | 17 | 14
Renal tubular necrosis (Renal and urinary disorders) | 19 | 17 | 20
Sinusitis (Infections and infestations) | 18 | 24 | 17
Tinea versicolour (Infections and infestations) | 15 | 11 | 6
Upper respiratory tract infection (Infections and infestations) | 52 | 56 | 60
Abdominal pain (Gastrointestinal disorders) | 40 | 48 | 47
Abdominal pain lower (Gastrointestinal disorders) | 6 | 13 | 13
Anaemia (Blood and lymphatic system disorders) | 86 | 92 | 85
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 54 | 51
C-reactive protein increased (Investigations) | 11 | 10 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 57 | 81 | 69
Diarrhoea (Gastrointestinal disorders) | 92 | 115 | 118
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 18 | 16
Ear pain (Ear and labyrinth disorders) | 3 | 13 | 5
Haemorrhoids (Gastrointestinal disorders) | 15 | 19 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 33 | 51 | 36
Mouth ulceration (Gastrointestinal disorders) | 3 | 7 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 27 | 19
Osteopenia (Musculoskeletal and connective tissue disorders) | 13 | 14 | 12
Pharyngitis (Infections and infestations) | 18 | 22 | 17
Pyrexia (General disorders) | 56 | 68 | 61
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 11
Weight decreased (Investigations) | 8 | 22 | 27
Abdominal distension (Gastrointestinal disorders) | 17 | 15 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 19 | 16
Candida infection (Infections and infestations) | 4 | 8 | 11
Complications of transplant surgery (Injury, poisoning and procedural complications) | 9 | 7 | 11
Decreased appetite (Metabolism and nutrition disorders) | 13 | 23 | 13
Dyslipidaemia (Metabolism and nutrition disorders) | 70 | 59 | 62
Erectile dysfunction (Reproductive system and breast disorders) | 14 | 8 | 10
Gout (Metabolism and nutrition disorders) | 11 | 10 | 2
Influenza (Infections and infestations) | 27 | 40 | 37
Leukocytosis (Blood and lymphatic system disorders) | 9 | 16 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 17 | 17
Nasopharyngitis (Infections and infestations) | 49 | 39 | 49
Neutropenia (Blood and lymphatic system disorders) | 10 | 14 | 9
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 11 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 28 | 19
Pneumonia (Infections and infestations) | 8 | 14 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 17 | 15
Urinary tract infection (Infections and infestations) | 77 | 91 | 71
Anxiety (Psychiatric disorders) | 27 | 26 | 27
Asthenia (General disorders) | 21 | 27 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 44 | 47
Cataract (Eye disorders) | 11 | 7 | 10
Chest pain (General disorders) | 21 | 17 | 22
Diabetes mellitus (Metabolism and nutrition disorders) | 15 | 19 | 23
Fatigue (General disorders) | 32 | 27 | 22
Hypercalcaemia (Metabolism and nutrition disorders) | 13 | 16 | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 12 | 9
Hypertrichosis (Skin and subcutaneous tissue disorders) | 11 | 0 | 4
Hypotension (Vascular disorders) | 31 | 36 | 45
Iron deficiency (Metabolism and nutrition disorders) | 8 | 11 | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 8 | 4
Oral candidiasis (Infections and infestations) | 14 | 11 | 19
Peripheral swelling (General disorders) | 9 | 8 | 12
Procedural pain (Injury, poisoning and procedural complications) | 40 | 40 | 41
Proteinuria (Renal and urinary disorders) | 30 | 41 | 30
Rash (Skin and subcutaneous tissue disorders) | 15 | 22 | 20
Tremor (Nervous system disorders) | 43 | 19 | 19
Aphthous ulcer (Gastrointestinal disorders) | 5 | 16 | 13
BK virus infection (Infections and infestations) | 11 | 9 | 13
Blood creatinine increased (Investigations) | 53 | 25 | 26
Chronic allograft nephropathy (Immune system disorders) | 21 | 4 | 5
Cytomegalovirus infection (Infections and infestations) | 19 | 13 | 10
Gastritis (Gastrointestinal disorders) | 12 | 14 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 20 | 19 | 19
Hyperuricaemia (Metabolism and nutrition disorders) | 36 | 11 | 8
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 4 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 11 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 9 | 16
Toxicity to various agents (Injury, poisoning and procedural complications) | 27 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.